# A Phase 2a, Randomized, Double-Blind Placebo-controlled, Parallel-group Study to Assess the Analgesic Efficacy and Safety of ASP8062 in Subjects with Fibromyalgia

## ISN/Protocol 8062-CL-0101

ClinicalTrials.gov Identifier: NCT03092726

Date of Statistical Analysis Plan v2.0: 19 Apr 2018

Sponsor: Astellas Pharma Global Development, Inc. (APGD)

1 Astellas Way Northbrook, IL 60062

# A Phase 2a, Randomized, Double-Blind Placebo-controlled, Parallel-group Study to Assess the Analgesic Efficacy and Safety of ASP8062 in Subjects with Fibromyalgia

## ISN/Protocol 8062-CL-0101

ClinicalTrials.gov Identifier: NCT03092726

Date of Statistical Analysis Plan v2.0: 19 Apr 2018

Sponsor: Astellas Pharma Global Development, Inc. (APGD)

1 Astellas Way Northbrook, IL 60062 ISN/Protocol 8062-CL-0101

### STATISTICAL ANALYSIS PLAN

Final Version 2.0, dated 19-Apr-2018

A Phase 2a, Randomized, Double-Blind Placebo-controlled, Parallel-group Study to Assess the Analgesic Efficacy and Safety of ASP8062 in Subjects with Fibromyalgia

ISN: 8062-CL-0101

IND number: 125639

Astellas Pharma Global Development, Inc. (APGD) 1 Astellas Way, Northbrook, IL 60062

\_\_\_\_\_

This confidential document is the property of the sponsor. No unpublished information contained in this document may be disclosed without prior written approval of the sponsor.

### **Table of Contents**

| I. | | LIS | T OF ABBREVIATIONS AND KEY TERMS······ 5 |
|---|---|---|---|
| 1 | | | TRODUCTION 9 |
| 2 | | FL | OW CHART AND VISIT SCHEDULE ······10 |
| 3 | | STU | UDY OBJECTIVE(S) AND DESIGN······15 |
| | 3.1 | | Study Objective(s) · · · · · 15 |
| | | 3.1.1 | Primary Objectives · · · · 15 |
| | | 3.1.2 | Secondary Objectives · · · · · 15 |
| | | 3.1.3 | 15 |
| | 3.2 | 2 | Study Design 15 |
| | 3.3 | | Randomization 16 |
| 4 | | SA | MPLE SIZE······16 |
| 5 | | AN | ALYSIS SETS ······17 |
| | 5.1 | | Full Analysis Set (FAS) · · · · · 17 |
| | 5.2 | 2 | Per Protocol Set (PPS) 17 |
| | | 5.2.1 | Reasons for Exclusion From PPS17 |
| | 5.3 | } | Safety Analysis Set (SAF) |
| | 5.4 | | Pharmacokinetics Analysis Set (PKAS) |
| 6 | | AN | ALYSIS VARIABLES ······20 |
| | 6.1 | | Efficacy Endpoints · · · · · · 20 |
| | | 6.1.1 | Primary Efficacy Endpoint(s) 20 |
| | | 6.1.2 | Secondary Efficacy Endpoints21 |
| | | 6.1.3 | 24 |
| | 6.2 | 2 | Safety Variables |
| | | 6.2.1 | Adverse Events · · · · 36 |
| | | 6.2.2 | Clinical Laboratory Variables |
| | | 6.2.3 | Vital Signs·····37 |
| | | 6.2.4 | Electrocardiograms ··········37 |
| | | 6.2.5 | Columbia Suicide Severity Rating Scale ··················37 |
| | 6.3 | 3 | Pharmacokinetic Variables 38 |
| | 6.4 | 1 | Other Variables · · · · 39 |
| | | 6.4.1 | Exposure39 |
| | | 6.4.2 | Percent Overall Compliance |

| | 6.4.3 | Previous and Concomitant Medication · · · · · 39 |
|---|---|---|
| | 6.4.4 | Time Since Onset of Fibromyalgia Symptoms and Time Since Diagnosis ······40 |
| | 6.4.5 | Mini-International Neuropsychiatric Interview ·······40 |
| | 6.4.6 | Widespread Pain Index and Symptom Severity Scale score ······40 |
| | 6.4.7 | Complex Medical Symptoms Inventory · · · · · 41 |
| | STA | ATISTICAL METHODOLOGY ······41 |
| 7. | .1 | General Considerations |
| 7. | .2 | Study Population ······43 |
| | 7.2.1 | Disposition of Subjects · · · · · 43 |
| | 7.2.2 | Protocol Deviations · · · · · 44 |
| | 7.2.3 | Demographic and Other Baseline Characteristics · · · · · 44 |
| | 7.2.4 | Previous and Concomitant Medications · · · · · 49 |
| | 7.2.5 | Previous and Concomitant Non-Medication Therapy50 |
| 7. | .3 | Study Drugs ······51 |
| | 7.3.1 | Exposure ······51 |
| | 7.3.2 | Treatment Compliance · · · · · 51 |
| 7. | .4 | Analysis of Efficacy |
| | 7.4.1 | Analysis of Primary Endpoint(s)52 |
| | 7.4.2 | Analysis of Secondary Endpoints · · · · · 55 |
| | 7.4.3 | 58 |
| | 7.4.4 | Analysis of Other Variables · · · · · 64 |
| 7. | .5 | Analysis of Safety 64 |
| | 7.5.1 | Adverse Events ······64 |
| | 7.5.2 | Adverse Events of Interest · · · · 65 |
| | 7.5.3 | Clinical Laboratory Evaluation · · · · · 66 |
| | 7.5.4 | Vital Signs·····68 |
| | 7.5.5 | Electrocardiograms ······70 |
| | 7.5.6 | Physical Examination Findings ······70 |
| | 7.5.7 | Columbia Suicide Severity Rating Scale · · · · · · · 70 |
| | 7.5.8 | Pregnancies 70 |
| 7. | .6 | Analysis of Pharmacokinetics70 |
| 7. | .7 | Analysis of Pharmacodynamics71 |
| 7. | .8 | Subgroups of Interest ······71 |
| | 7.8.1 | Subgroup Analysis for Primary Endpoint ······71 |

| | | 7.8.2 | 72 |
|---|---|---|---|
| | 7.9 | ) ( | Other Analyses · · · · · · · 72 |
| | 7.1 | l0 I | nterim Analysis (and Early Discontinuation of the Clinical Study) ·······73 |
| | 7.1 | 1 F | Handling of Missing Data, Outliers, Visit Windows, and Other Information ······73 |
| | | 7.11.1 | Missing Data · |
| | | 7.11.2 | Outliers76 |
| | | 7.11.3 | Values Below Limit of Quantification (BLOQ) · |
| | | 7.11.4 | Visit Windows for Efficacy Variables · |
| | | 7.11.5 | Visit Windows for Safety Variables · · · · · · · 78 |
| | | 7.11.6 | Pooling Sites Algorithm · · · · · 80 |
| 8 | | DOC | UMENT REVISION HISTORY ····· 80 |
| 9 | | REFI | ERENCES87 |
| 10 | | APPE | ENDICES88 |
| | 10. | .1 A | Appendix 1: Drug Abuse Related Adverse Events······88 |
| | 10. | .2 A | Appendix 2: Drug Withdrawal Related Adverse Events · · · · · · 91 |
| | 10. | .3 A | Appendix 3: Potentially Clinically Significant Laboratory Criteria93 |
| | 10. | .4 <i>A</i> | Appendix 4: Key Contributors and Approvers ······94 |

### I. LIST OF ABBREVIATIONS AND KEY TERMS

#### **List of Abbreviations**

| Abbreviations | Description of abbreviations |
|---|---|
| ACR | American College of Rheumatology |
| AE | Adverse Event |
| ALP | Alkaline Phosphatase |
| ALT | Alanine Transaminase |
| ANCOVA | Analysis of Covariance |
| ANOVA | Analysis of Variance Analysis of Variance |
| APGD | Astellas Pharma Global Development, Inc. |
| ASCM | |
| | Analysis Set Classification Meeting |
| AST | Aspartate Transaminase |
| ATC | Anatomical Therapeutic Chemical |
| BLOQ | Below the Limit of Quantification |
| BMI | Body Mass Index |
| BOCF | Baseline Observation Carried Forward |
| CI | Confidence Interval |
| CMSI | Complex Medical Symptom Inventory |
| CSR | Clinical Study Report |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| DBP | Diastolic Blood Pressure |
| DSM-V | Diagnostic and Statistical Manual of Mental Disorders |
| e-diary | Electronic diary |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| EOS | End of Study |
| EOT | End of Treatment |
| EQ-VAS | EQ Visual Analog Scale |
| FAS | Full Analysis Set |
| FIQR | Fibromyalgia Impact Questionnaire Revised |
| FM | Fibromyalgia |
| FU | Follow-up |
| GD-US | Global Development - United States |
| Н | High |
| HADS | Hospital Anxiety and Depression Scale |
| IAP | Interim Analysis Plan |
| ICD-10 | International Statistical Classification of Diseases and Related Health Problems |
| ICF | Informed Consent Form |
| ICH | International Council for Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDIVIC | macpendent Data Womtoring Committee |

| Abbreviations | Description of abbreviations |
|---------------|-----------------------------------------------|
| INR | International Normalized Ratio |
| IRT | Interactive Response Technology |
| L | Low |
| LDH | Lactate Dehydrogenase |
| LOCF | Last Observation Carried Forward |
| LS | Least Squares |
| mBOCF | Modified Baseline Observation Carried Forward |
| MDD | Major Depressive Disorder |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | Multiple Imputation |
| M.I.N.I. | Mini-International Neuropsychiatric Interview |
| MMRM | Mixed Model Repeated Measures |
| N | Normal |
| NRS | Numerical Rating Scale |
| NSAID | Nonsteroidal Anti-inflammatory Drug |
| PCS | Potentially Clinically Significant |
| PD | Protocol Deviation |
| PGIC | Patient Global Impression of Change |
| PGIS | Patient Global Impression of Severity |
| PK | Pharmacokinetic |
| PKAS | Pharmacokinetics Analysis Set |
| PPS | Per-Protocol Analysis Set |
| PRO | Patient Reported Outcome |
| PT | Preferred Term |
| RBC | Red Blood Cell |
| SAE | Serious Adverse Event |
| SAF | Safety Analysis Set |
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analysis Software |
| SBP | Systolic Blood Pressure |
| SD | Standard Deviation |
| SE | Standard Error |
| SMQ | Standardized MedDRA Query |
| SOC | System Organ Class |
| SS | Symptom Severity |
| TBL | Total Bilirubin |
| TEAE | Treatment Emergent Adverse Event |
| THC | Tetrahydrocannabinol |

| Abbreviations | Description of abbreviations |
|---------------|-------------------------------------------|
| TLF | Tables, Listings and Figures |
| ULN | Upper Limit of Normal |
| US | United States |
| WBC | White Blood Cell |
| WHO-DD | World Health Organization Drug Dictionary |
| WPI | Widespread Pain Index |

### **List of Key Terms**

| Terms | Definition of terms |
|---|---|
| Baseline Diary Run-In | 7-day period in which subject completes numerical rating scale (NRS) on handheld device daily beginning at Day -7 through Day -1. |
| End of Study | End of study for each subject has occurred when the final protocol-defined assessment has been completed. In this study, the last protocol defined assessment is approximately 4 weeks after last study drug dose. |
| End of Treatment | The date the last dose of study drug was taken by the enrolled subject. |
| Randomization | The process of assigning trial subjects to treatment or control groups using an element of chance to determine assignments in order to reduce bias. Randomization will occur after predose assessments and eligibility criteria have been confirmed at Visit 3. |
| Treatment-Emergent<br>Adverse Event | Any adverse event which starts, or worsens, after the first dose of study drug through 30 days after the last dose of study drug. |

ISN/Protocol 8062-CL-0101

#### 1 INTRODUCTION

This Statistical Analysis Plan (SAP) contains a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and includes detailed procedures for executing the statistical analysis of the primary and secondary endpoints and other data.

The SAP is finalized and signed prior to database hard lock to ensure lack of bias. Any subsequent changes will be described with justification in an updated version of the SAP (with date of version number).

This statistical analysis is coordinated by the responsible biostatistician of GD-US. Any changes from the analyses planned in the SAP will be justified in the Clinical Study Report (CSR).

Prior to database hard lock, a final review of data and Tables, Listings and Figures (TLFs) meeting will be held to allow a review of the clinical trial data and to verify the data that will be used for analysis set classification. If required, consequences for the statistical analysis will be discussed and documented. A meeting to determine analysis set classifications may also be held prior to database hard lock.

#### 2 FLOW CHART AND VISIT SCHEDULE

Figure 1 Study flow chart



| Visit Day: -42 | -7 | 1 | 15 | 29 | 57 | 71 | 85 |
|----------------------|----|---|----|----|----|----|----|
| Visit Week: -6 to -1 | -1 | | 2 | 4 | 8 | 10 | 12 |

EOS: end of study; EOT: end of treatment.

 Table 1
 Schedule of Assessments

| | So | creening Perio | d | | , | Treatment Per | Follow-Up Period <sup>a</sup> | | |
|---|---|---|---|---|---|---|---|---|---|
| Schedule of Assessments | Screening Wash-out | | Baseline<br>Diary<br>Run-In | Randomization | Treatment | | | Follow-up<br>Visit | End of Study<br>(EOS)<br>Phone Call |
| Visit | 1 | NA | 2 | 3 | 4 | 5 | 6 | 7 | N/A |
| Week | | -6 through -1 | | | 2 | 4 | 8/EOT | 10 | 12 |
| Day (and Window) | -42 1 | to -8 | -7 to -1 | 1 | $15 \pm 2$ | $29 \pm 2$ | $57 \pm 2$ | $71 \pm 2$ | $85 \pm 2$ |
| ASSESSMENTS | | | | | | | | | |
| Informed Consent | X | | | | | | | | |
| Demographics | X | | | | | | | | |
| Height and Weight <sup>b</sup> | X | | | X | | X | X | | |
| Medical/Surgical History | X | | X <sup>c</sup> | | | | | | |
| Medication History and | X | | | | | | | | |
| Concomitant Medication | Λ | | | | | | | | |
| FM Diagnosis (ACR 1990 & 2010) | X | | | | | | | | |
| Verify Eligibility Criteria (and | X | $X^d$ | X <sup>d</sup> | X | | | | | |
| duplicate subject database check) | Λ | | Λ | Λ | | | | | |
| Phone Call to Subject <sup>e</sup> | | X | | | | | | | X |
| e-diary Distribution/Return | | | X | | | | | X | |
| Physical Examination (including | X | | | X | | | X | X | |
| tender point exam at screening) | | | | | | | Λ | Λ | |
| Drug and Alcohol Screen <sup>f</sup> | X | | X | X | | | | | |
| Randomization <sup>g</sup> | | | | X | | | | | |
| Vital Signs <sup>h</sup> | X | | | X | X | X | X | X | |
| Laboratory Tests (Hematology, | X | | | X | X | X | X | X | |
| Biochemistry, Urinalysis) <sup>i</sup> | | | | | Λ | Λ | | | |
| Electrocardiogram <sup>j</sup> | X | | | X | | | X | X | |
| Pregnancy Test | $X^k$ | | | X <sup>l</sup> | | | $X^{l}$ | X <sup>l</sup> | |
| Blood Sample for | | | | X | | | | | |
| Pharmacogenomics <sup>m</sup> | | | | Λ | | | | | |
| Blood sampling for | | | | X | X | X | X | | |
| Pharmacokinetics <sup>n</sup> | | | | Λ | Λ | Λ | Λ | | |
| Table continued on next page | | | | | | | | | |

| | Screening Period | | | | | Treatment Per | Follow-Up Period <sup>a</sup> | | |
|---|---|---|---|---|---|---|---|---|---|
| Schedule of Assessments | Screening | Wash-out | Baseline<br>Diary<br>Run-In | Randomization | Treatment | | Follow-up<br>Visit | End of Study<br>(EOS)<br>Phone Call | |
| Visit | 1 | NA | 2 | 3 | 4 | 5 | 6 | 7 | N/A |
| Week | | -6 through -1 | | | 2 | 4 | 8/EOT | 10 | 12 |
| Day (and Window) | -42 | to -8 | -7 to -1 | 1 | $15 \pm 2$ | 29 ± 2 | $57 \pm 2$ | $71 \pm 2$ | $85 \pm 2$ |
| CMSI | | | X | | | | | | |
| MINI° | X | | | | | | | | |
| HADS <sup>p</sup> | X | | | X | | | X | | |
| NRS e-diary Collection <sup>q</sup> | | | $\leftarrow$ | _ | | | | $\longrightarrow$ | |
| PGICs | | | | | X | X | X | X | |
| PGIS <sup>t</sup> | | | | X | X | X | X | X | |
| | | | | | | | | _ | |
| | | | | | _ | _ | | | |
| | | | $\leftarrow$ | | | | | $\rightarrow$ | |
| FIQR <sup>x</sup> | X | | | X | X | X | X | X | |
| C-SSRS | X | | | X | X | X | X | X | |
| Subject Training Materials <sup>aa</sup> | X | | X | | | | | | |
| Study Drug Dispensed | | | | X | X | X | | | |
| Study Drug Dosingbb | | | | X | X | X | X | | |
| Study Drug Returned | | | | | X | X | X | | |
| Adverse Events <sup>cc</sup> | < | | | | | | | | $\longrightarrow$ |
| Rescue Medication (if applicable) | | | <del></del> | | | | | $\longrightarrow$ | |

- a) Follow-up visit and phone call will be planned relative to date of last dose (14 and 28 days post last dose).
- b) Height will be measured at screening only. Weight will be collected at screening, prior to randomization, week 4 and week 8/BOT.
- c) Any change between the screening and randomization visits will also be captured in the medical/surgical history.
- d) Continued subject eligibility to be confirmed based on laboratory results prior to having the subject wash-out of current pain medications (phone call). Continued subject eligibility to be confirmed based on completion of wash-out prior to having the subjects start baseline diary run-in (visit 2).

Footnotes continued on next page

- e) During screening period (wash-out): Study staff to contact the subject, if necessary, to initiate wash-out of current pain medications after continued eligibility has been confirmed. During follow up: Follow-up phone call 4 weeks (day 85) post study drug will be required.
- f) Subjects will be tested for drugs and alcohol at screening, baseline diary run-in and randomization. A positive test for tetrahydrocannabinol (THC) and/or opioids is allowed at the screening visit, but must be confirmed negative prior to baseline diary run-in and randomization.
- g) Continued subject eligibility to be assessed and confirmed based on daily average pain scores recorded in the e-diary prior to subject being randomized.
- h) Resting blood pressure and pulse rate values will be the average of the supine triplicates from the orthostatic measures for those days when orthostatic blood pressure is assessed. Pulse rate will be measured in triplicate after the subject has rested for at least 7 minutes in the supine position, each measurement approximately 1 minute apart (-3, -2, and -1 minutes before standing). Afterwards, the subject will be instructed to stand up within 10 seconds and remain free standing with no support on wall or furniture. Standing blood pressure and pulse rate will be measured after the subject has been in the free standing position at 3 minutes (every attempt should be made to take the measurement as close as possible to 3 minutes). Orthostatic vital signs will be captured on day 1 pre-dose and approximately 2 hours post dose and at week 8/EOT. Resting vital sign measurements should be conducted prior to blood draws. Body temperature will be assessed at screening, randomization and week 8/EOT only.
- i) Blood specimens for scheduled clinical chemistry laboratory tests do not need to be fasted samples.
- j) Electrocardiograms are to be conducted prior to blood draws. A single electrocardiogram (ECG) will be obtained at the specified visits, unless, in the investigator's judgment, additional ECG's are required for safety reasons.
- k) Serum for females of childbearing potential.
- 1) Urine for females of childbearing potential. Sample is to be collected prior to randomization, and at week 8/EOT, and week 10/ follow-up visits.
- m) Sample to be collected one time, preferably prior to first dose on day 1; however, can be collected at any time during the course of the study. Separate pharmacogenomics informed consent will need to be obtained from subject prior to collecting.
- n) A single pharmacokinetic sample will be taken on day 1 in the clinic at approximately 1-4 hour(s) after dosing and once at each visit during weeks 2, 4 and 8/EOT. PK samples at weeks 2, 4, and 8/OT should be evenly split between the following 3 sampling windows: before dosing, 1-4 hours post dose and >4 hours post dose. Time of the last dose and time of sample collection will be captured in the eCRF during these visits.
- o) Mini-International Neuropsychiatric Interview (MINI) will be completed by site personnel at screening.
- p) Hospital Anxiety and Depression Scale (HADS). Questionnaire will be completed by the subject at screening, randomization and the week 8/EOT visits.
- q) Numeric Rating Scale (NRS). Subject is to rate average pain on a daily basis (24 hour recall) by entering pain score (0 10) in the e-diary. The NRS should be completed prior to bedtime at a consistent time of day throughout the study starting daily at diary run-in until week 10.
- s) Patient Global Impression of Change (PGIC). Questionnaire will be completed by the subject at week 2, 4 and 8/EOT follow-up visits.
- t) Patient Global Impression of Severity (PGI-S). Questionnaire will be completed by the subject at randomization and week 2, 4 and 8/EOT follow-up visits.
- $\mathbf{u}$ )
- Footnotes continued on next page

r)

v)

w)

x) Fibromyalgia Impact Questionnaire Revised (FIQR) will be completed by the subject at screening, randomization and at week 2, 4, 8/EOT and week 10/follow up visits. At screening, subject only completes the item for pain of the FIQR.

v)

- z) Columbia Suicide Severity Rating Scale (C-SSRS). Questionnaire will be facilitated by the Principal Investigator/Site staff, as appropriately trained, at screening, randomization, weeks 2, 4, 8/EOT, and week 10/follow up visits.
- aa) Subject Training Materials are to be distributed and reviewed during the screening period.
- bb) Subjects will begin study drug dosing on day 1 of the randomization visit.
- cc) (Serious) Adverse Events will be collected from the time of signing the informed consent through 4 weeks post-last dose.

19-Apr-2018 Astellas Page 14 of 96

ISN/Protocol 8062-CL-0101

### 3 STUDY OBJECTIVE(S) AND DESIGN

### 3.1 Study Objective(s)

The objectives of the study, conducted in subjects with fibromyalgia, are the following:

#### 3.1.1 Primary Objectives

- Assess analgesic efficacy of ASP8062 relative to placebo.
- Assess the safety and tolerability of ASP8062 relative to placebo.

#### 3.1.2 Secondary Objectives

- Assess treatment differences in physical function of ASP8062 relative to placebo.
- Assess the improvements in overall subject status (e.g., fibromyalgia symptoms, global functioning) of ASP8062 relative to placebo.



# 3.2 Study Design

This is a Phase 2a, randomized, double-blind, placebo-controlled parallel group study to assess analgesic efficacy and safety of ASP8062 in subjects with fibromyalgia.

The study will be conducted in the United States (US) in up to 35 sites. Approximately 356 subjects are planned to be screened for 178 randomized subjects (89/arm; 50% screen fail rate). Subjects will be randomized in a 1:1 ratio to one of two treatment groups: ASP8062 30 mg or Placebo once per day.

The study will consist of a screening period of up to 6 weeks, which includes the completion of screening procedures, wash-out of prohibited medications (if applicable) followed by a 1-week baseline diary run-in; an 8-week double-blind randomized treatment period (subjects randomized to the ASP8062 group will receive ASP8062 30 mg [1 tablet of 25 mg and 1 tablet of 5 mg] once daily; subjects randomized to the placebo group will receive placebo [2 tablets] to match ASP8062 once daily); and a 4-week follow-up period. The total study duration for a subject is approximately 18 weeks.

Acetaminophen may be used as rescue therapy for intolerable pain due to fibromyalgia during the baseline diary run-in and in all subsequent study periods. Nonsteroidal

anti-inflammatory drugs (NSAIDs) may be used (with the exception of celecoxib) as needed for non-fibromyalgia pain (e.g., headache). Subjects are encouraged to abstain from alcohol.

This study design includes a stopping rule for futility. Two interim analyses for futility based on the primary efficacy endpoint will be conducted. The timing of these analyses will be at approximately 35% and 55% of all subjects with Week 8/End of Treatment (EOT) data. The plan for the interim analysis may be modified based on speed of recruitment.

The futility analyses will be conducted by an Astellas statistician, with results reviewed by an Astellas Independent Data Monitoring Committee (IDMC). The Astellas statistician and other members of the Astellas IDMC are external to the study team. No one within the study team will be unblinded to the treatment allocation or interim results. Details of the interim analysis procedure, steps to maintain treatment blind in the study team and criteria for stopping the study will be described in an Interim Analysis Plan (IAP).

#### 3.3 Randomization

All subject numbers will be assigned using the interactive response technology (IRT) starting at screening. All subjects will have a unique, ten-digit subject number. The first five digits of this number will be the investigator's site number. The second five digits assigned will represent the subject's accession number. This will be the number that identifies a subject during the course of the study.

Screening procedures, wash-out of prohibited medications (if applicable) and the baseline-diary run-in will be completed prior to randomization. Only subjects who meet all inclusion criteria and exhibit none of the exclusion criteria will be randomly assigned in a 1:1 ratio to ASP8062 30 mg or placebo according to the randomization schedule through IRT. The randomization will be stratified by site. Site personal will dispense the treatment according to the IRT system's assignment.

If a subject is assigned a randomization number, but does not receive study drug, the randomization number will not be used again.

The randomization schedules that determine subject treatment will be computer-generated by IRT before the beginning of the study. Specific procedures for randomization through the IRT are contained in the study-specific IRT manual.

#### 4 SAMPLE SIZE



ISN/Protocol 8062-CL-0101



#### 5 ANALYSIS SETS

In accordance with International Council for Harmonization (ICH) recommendations in guidelines E3 and E9, the following analysis sets will be used for the analyses.

Detailed criteria for analysis sets will be laid out in Classification Specifications and for the allocation of subjects to analysis sets, except Pharmacokinetic Analysis Set (PKAS), will be determined prior to database hard lock. The allocation of subjects to PKAS will be determined after database hard lock.

### 5.1 Full Analysis Set (FAS)

The full analysis set (FAS) will consist of all randomized subjects who take at least one dose of study drug.

The FAS will be used for demographic and baseline characteristic summaries and primary summaries and analyses of efficacy variables.

When the FAS is utilized in an analysis, subjects will be presented by the randomized treatment group, i.e. planned treatment group, even if the treatment they received was different.

# 5.2 Per Protocol Set (PPS)

The per protocol set (PPS) will include a subset of subjects from the FAS who meet criteria based on adherence to the protocol, which may affect the primary efficacy endpoint or select secondary efficacy endpoints. The PPS criteria is defined in Section 5.2.1 of this SAP.

The PPS will be used for demographic and baseline characteristic summaries and for sensitivity analyses of the primary endpoint and select secondary efficacy endpoints outlined in Section 7.4.2

Final judgments on exclusion of subjects from the PPS are to be made at the analysis set classification meeting (ASCM), which will be held prior to database hard lock and unblinding of the study.

#### 5.2.1 Reasons for Exclusion From PPS

A subject who meets any of the criteria described in Table 2 will be completely excluded from the PPS; there will be no partial data exclusion of a specified time point for a subject.

 $\textbf{Sponsor:} \ Astellas \ Pharma \ Global \ Development, \ Inc. \ (APGD)$ 

ISN/Protocol 8062-CL-0101

**Table 2** Criteria for Assessing Reasons for Exclusion From PPS

| Number | Source | Criterion/Criteria |
|---|---|---|
| Didn't Sat | isfy Diary Eligibility Criteria | |
| 1.1 | Inclusion Criterion # 13: Subject is compliant with daily pain recordings during the baseline diary run-in period, as defined by the completion of a minimum of 5 of 7 daily average pain ratings. | Compliance is not met at baseline i.e. number of days of daily average NRS pain ratings during the baseline diary run-in (from study day -7 to -1) is < 5 |
| 1.2 | Inclusion Criterion # 14: Subject has a mean daily average pain score ≥ 4 and ≤ 9 on an 11 point 0 to 10 NRS as recorded in the subject electronic diary (e-diary) during the baseline diary run-in period, and meeting pre-specified criteria for daily average pain scores. | <ul> <li>During the baseline diary run-in period (from study day -7 to -1) the subject has:</li> <li>A mean daily average pain NRS of &lt; 4 or &gt; 9 and/or,</li> <li>Two or more daily average pain scores of &gt; 9 and/or,</li> <li>Four or more daily average pain scores of ≤ 3.</li> </ul> |
| Didn't Sat | isfy Non-Diary Eligibility Criteria | |
| 2.1 | <ul> <li>Inclusion Criterion # 10:</li> <li>Subject meets the American College of Rheumatology (ACR) 1990 fibromyalgia diagnostic criteria at Screening: <ul> <li>Widespread pain for at least 3 months, defined as the presence of all of the following: <ul></ul></li></ul></li></ul> | Inclusion Criterion # 10 is No and/or pain in <11 tender point sites |
| 2.2 | <ul> <li>Inclusion Criterion # 11:</li> <li>Subject meets the ACR 2010 fibromyalgia diagnostic criteria at Screening:</li> <li>Widespread pain index (WPI) ≥ 7 and symptom severity (SS) scale score ≥ 5 or WPI 3-6 and SS scale score ≥ 9.</li> <li>Symptoms have been present at a similar level for at least 3 months.</li> <li>The subject does not have a disorder that would otherwise explain the pain.</li> </ul> | Inclusion criterion #11 is No and/or<br>WPI >=7 and SS scale score <5 or<br>WPI 3-6 and SS scale <9 or<br>WPI<3 |
| 2.3 | Inclusion Criterion # 12: Subject has a pain score ≥ 4 on the revised fibromyalgia impact questionnaire revised (FIQR) pain item at Screening. inued on next page | Inclusion criterion #12 is No and/or FIQR pain item score <4 at Screening. |

| Number | Source | Criterion/Criteria |
|---|---|---|
| | sion Criteria | |
| 3.1 | Exclusion Criterion # 4: Subject has pain due to diabetic peripheral neuropathy, post-herpetic neuralgia, traumatic injury, prior surgery, complex regional pain syndrome, or other source of pain that, in the investigator's opinion, would confound or interfere with the assessment of the subject's fibromyalgia pain or require excluded therapies during the subject's study participation. Exclusion Criterion # 5: | Exclusion Criterion # 4 is Yes. Exclusion Criterion # 5 is Yes. |
| 3.2 | Subject has infectious or inflammatory arthritis (e.g., rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis and gout), autoimmune disease (e.g., systemic lupus erythematosus), or other widespread rheumatic disease other than fibromyalgia. | Exclusion Citerion # 3 is 1es. |
| 3.3 | Exclusion Criterion # 6: Subject has a current, untreated moderate or severe major depressive disorder (MDD) as assessed by the Mini-International Neuropsychiatric Interview (M.I.N.I.). Subject with current, treated major depressive disorder can be included provided that, in the investigator's opinion, it is without clinically significant changes in symptoms while on the same dose of a protocol allowed antidepressant for greater than 60 days prior to Screening. | Exclusion Criterion # 6 is Yes. |
| 3.4 | Exclusion Criterion # 8:<br>Subject has a history of any psychotic and/or<br>bipolar disorder as assessed by the M.I.N.I. | Exclusion Criterion # 8 is Yes. |
| 3.5 | Exclusion Criterion # 9:<br>Subject has a HADS score > 14 on the Depression<br>subscale at Screening or at the time of Visit 3<br>(Randomization). | HADS Depression subscale score > 14 at Screening or Visit 3 (Randomization), or Exclusion Criterion #9 is Yes. |
| Error in S | tudy Drug Administration Compared to Treatment | |
| 4 | Received wrong treatment during the double-blind treatment period | A subject will be excluded if the study drug taken at any time during the double-blind treatment period is different from the treatment group assigned at randomization. |
| Poor Stud | y Drug Compliance | 1 |
| 5 | Poor study drug compliance during the double-blind treatment period. | Percent overall compliance is <70% for a subject, calculated over Study Day 1 to Week 8/EOT. Subjects with missing compliance will be reviewed on a case-by-case basis. |
| Table cont | inued on next page | |

| Number | Source | Criterion/Criteria |
|---|---|---|
| Unblinding of Study Drug | | |
| 6 | Incorrect unblinding of double-blind study drug. | A subject's treatment for double-blind study drug is incorrectly unblinded. The decision to exclude the subject will be evaluated on a case by case basis. |
| Use of Prohibited Concomitant Medication | | |
| 7 | Subject received celecoxib, duloxetine, gabapentin, milnacipran or pregabalin, during the double-blind treatment period. | Subject received at least one dose of received celecoxib, duloxetine, gabapentin, milnacipran or pregabalin during the double-blind treatment period. |

# 5.3 Safety Analysis Set (SAF)

The Safety Analysis Set (SAF) consists of all randomized subjects who received at least one dose of study drug.

The SAF will be used for summaries of demographic and baseline characteristics and all safety and tolerability related variables.

When the SAF is utilized in an analysis, subjects will be presented by the treatment actually received. Subjects who are randomized to placebo who accidentally receive at least one dose of ASP8062 will be summarized in the ASP8062 treatment group in the SAF.

### 5.4 Pharmacokinetics Analysis Set (PKAS)

The PKAS will consist of the subset of SAF for which at least one post dose concentration is available.

#### 6 ANALYSIS VARIABLES

# **6.1** Efficacy Endpoints

The subjects will use a handheld device (an e-diary that will be taken home) to report daily average pain NRS scores, and to capture rescue medication use. Data will be automatically transmitted to a central database.

The questionnaires on efficacy to be performed during the clinic visits (Fibromyalgia Impact Questionnaire Revised [FIQR], Patient Global Impression of Change [PGIC], Patient Global Impression of Severity [PGIS],

Ind Hospital Anxiety and Depression

Scale [HADS]) depression subscale will be reported on a tablet device that is available at the site. For FIQR, PGIS, and HADS, baseline is defined as the last assessment on or prior to the first dose day (Day 1) of double-blind study drug.

#### 6.1.1 Primary Efficacy Endpoint(s)

The primary efficacy variable is the change from baseline to Week 8 in mean daily average pain score assessed by NRS (0 to 10 scale).

The NRS is a generic instrument for the assessment of pain, consisting of a single question that asks subjects to record their daily average pain on an 11- point scale, where 0 anchors "no pain" and 10 "pain as bad as you can imagine." The recall period is the last 24 hours.

The subject will use the e-diary to report daily average pain NRS scores from the start of the baseline diary run-in period through Week 10. Subjects will be instructed to complete the NRS in the evening and at a consistent time each day (ideally between 6pm and midnight, however can be captured until 2am the next morning). For this reason, any daily average pain score entered onto the e-diary up to 2am the following day will be attributed to the previous study day in the derivation of the mean daily average NRS pain scores. This is described in more detail in Section 7.11.4.3

Mean daily average NRS pain scores will be derived for each subject as follows:

Table 3 Derivation of mean daily average NRS pain score

| <b>Analysis Time Point</b> | Derivation |
|---|---|
| Baseline | Arithmetic mean of non-missing daily pain scores from the last 7 days prior to the randomization visit i.e., using the non-missing scores from Study Days -7 to -1. If the pain score is missing on all of these 7 days, then the score will be set to missing. |
| Treatment period Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, EOT | Arithmetic mean of non-missing daily pain scores collected within time window per visit windows defined in Section 7.11.4.3 Table 26 If the pain score is missing on all of the days during the time window, then the score for that time point will be set to missing. |
| Follow-up period<br>Week 10 | |

EOT: end of treatment

Change from baseline is defined in Section 7.1 A negative change indicates a reduction/improvement from baseline (i.e., a favorable outcome).

#### **6.1.2** Secondary Efficacy Endpoints

Secondary efficacy endpoints include:

- Percentage of subjects achieving ≥ 30 % (or ≥ 50%) reduction from baseline to Week 8 in mean daily average pain score assessed by NRS (0 to 10 scale) in the subject's daily diary.
  - A subject with at least 30% (or 50%) reduction in mean daily average pain score (NRS) from baseline to Week 8 will be classified as a responder; otherwise they will be classified as a non-responder.
  - o Subjects who do not have Week 8 data will be classified as non-responders.
  - o Subjects who do not have baseline data will be classified as non-responders.
- Percentage of subjects achieving  $\geq 30$  % (or  $\geq 50$ %) reduction from baseline to EOT in mean daily average pain score assessed by NRS (0 to 10 scale) in the subject's daily diary.

- A subject with at least 30% (or 50%) reduction in mean daily average pain score (NRS) from baseline to EOT will be classified as a responder; otherwise they will be classified as a non-responder.
- Subjects who do not have EOT data will be classified as non-responders.
- o Subjects who do not have baseline data will be classified as non-responders.

Percent change from Baseline is defined in Section 7.1 A negative percent change indicates a reduction/improvement from Baseline (i.e., a favorable outcome).

• Change from baseline to Weeks 2, 4, 8 and EOT in the FIQR function, symptoms and overall impact subscales.

The 21-item FIQR contains 3 subscales: function (9 questions), overall impact (2 questions), and symptoms (10 questions). Subjects answer each question on an 11-point NRS, with anchors appropriate to each question on a tablet device during the clinic visit. The recall period is the last 7 days or, for the function subscale, the last time the activity was performed if not within the 7-day recall period.

For each subject the items described in <u>Table 4</u> will be derived. The questionnaire should be considered to be invalid if three or more of the individual questions are unanswered. In this case, all subscales and the total score would be set to missing, even if a particular subscale has no missing items.

Change from baseline is defined in Section 7.1 A negative change indicates a reduction/improvement from baseline (i.e., a favorable outcome).

Table 4 Derivation of FIQR Subscales and Total Score

| Analysis Time | FIQR Item | Derivation |
|---|---|---|
| Point | | |
| Baseline, | Function subscale score Rate the difficulty of the following | Sum of scores from questions 1 to 9. |
| Treatment period | activities: | In the case of missing data, unanswered |
| Week 2, Week 4, | 3) Brush or comb your hair | questions should be compensated using the |
| Week 8, EOT, | 4) Walk continuously for 20 mins | following "weighting" factor: |
| | 5) Prepare a homemade meal | If only x questions from the Function |
| Follow-up period | 6) Vacuum, scrub or sweep floors | subscale were answered, the added score of |
| Week 10 | 7) Lift and carry a full bag of groceries | the x questions should be weighed by 9/x. |
| | 8) Climb one flight of stairs | The range of scores will be 0 to 90, with a |
| | 9) Change bed sheets | lower score indicting better (higher) |
| | 10) Sit in a chair for 45 mins | function. |
| | 11) Go shopping for groceries | |
| | Overall impact subscale score: | Sum of scores from questions 10 and 11. |
| | <ul><li>12) Fibromyalgia prevented me from accomplishing goals for the week</li><li>13) I was completely overwhelmed by my fibromyalgia symptoms</li></ul> | In the case of missing data, unanswered questions should be compensated using the following "weighting" factor: If only x questions from the Overall impact subscale were answered, the added score of the x questions should be weighed by 2/x. |
| | | The range of scores will be 0 to 20, with a lower score indicating better (lower) impact. |
| | Symptoms subscale score: | Sum of scores from questions 12 to 21. |
| | Please rate: | duni er seeres from questions 12 to 21. |
| | 14) Your level of pain | In the case of missing data, unanswered |
| | 15) Your level of energy | questions should be compensated using the |
| | 16) Your level of stiffness | following "weighting" factor: |
| | 17) The quality of your sleep | If only x questions from the Symptoms |
| | 18) Your level of depression | subscale were answered, the added score of |
| | <ul><li>19) Your level of memory problems</li><li>20) Your level of anxiety</li></ul> | the x questions should be weighed by 10/x. |
| | <ul><li>21) Your level of tenderness to touch</li><li>22) Your level of balance problems</li><li>23) Your level of sensitivity to loud noises, bright lights, odors and colds</li></ul> | The range of scores will be 0 to 100, with a lower score indicating a better (lower) level of symptoms. |
| | Total score | A normalization factor is applied to each of the three subscale scores: the function subscale score is divided by 3, the overall subscale score is divided by 1 (i.e. it is left unchanged), and the symptoms subscale score is divided by 2. |
| | | The total FIQR score is the sum of the three normalized subscale scores. The range of scores will be 0 to 100, with a lower score indicating a better response. |

EOT: end of treatment

• Overall subject improvement assessed by PGIC at Weeks 2, 4, 8, and EOT.

The PGIC is a self-administered 7-point Likert scale that asks subjects to evaluate their fibromyalgia relative to baseline. This is a single question and the grade ranges from 1 to 7, where 1 anchors "Very Much Improved" and 7 anchors "Very Much Worse". Subjects will complete the questionnaire during the clinic visits on a tablet device.
























# The schedule of safety assessments is shown in Table 1 Baseline is defined as the last assessment on or prior to the first dose day (Day 1) of double-blind study drug.

## **6.2.1** Adverse Events

Adverse events will be categorized as those which occur prior to first dose or treatment-emergent as follows:

- Adverse events prior to first dose
  Adverse events prior to first dose is an adverse event which starts prior to the first dose
  of study drug. If the adverse event occurs on Day 1 and the onset check box is marked
  "Onset before first dose of study drug", then the adverse event will be considered as an
  AE prior to first dose. If the adverse event occurs on Day 1 and the onset check box is
  marked "Onset after first dose of study drug" or the onset check box is left blank, then
  the adverse event will not be considered as an AE prior to first dose.
- Treatment-emergent adverse events (TEAEs; frequency, severity, seriousness, and relationship to study drug).

<u>TEAE</u> is defined as an adverse event which starts, or worsens, after the first dose of study drug through 30 days after the last dose of study drug. If the adverse event occurs on Day 1 and the onset check box is marked "Onset after first dose of study drug" or the onset check box is left blank, then the adverse event will be considered treatment emergent. If the adverse event occurs on Day 1 and the onset check box is marked "Onset before first dose of study drug", then the adverse event will not be considered treatment emergent, unless it worsens in severity after Day 1 (up to day 30 after last dose).

<u>TEAE (Treatment period)</u> is an adverse event which starts, or worsens, after the first dose of study drug through to 4 days after the last dose of study drug. If the adverse event occurs on Day 1 and the onset check box is marked "Onset after first dose of study drug" or the onset check box is left blank, then the adverse event will be considered treatment emergent. If the adverse event occurs on Day 1 and the onset check box is marked "Onset before first dose of study drug", then the adverse event will not be considered treatment emergent, unless it worsens in severity after Day 1 (up to day 4 after last dose).

<u>TEAE (Follow-up period)</u> is an adverse event which starts, or worsens, 5 days after the last dose of study drug through 30 days after the last dose of study drug.

<u>A drug-related TEAE</u> is defined as any TEAE with a possible or probable relationship to study treatment as assessed by the investigator or with missing assessment of the causal relationship.

For each AE, duration will be calculated in days, using the following formula:

• Duration of AE = End date of AE - Start date of AE +1,

where the start <u>date of AE</u> and the end <u>date of AE</u> are defined as the onset date and end date of the AE, as captured in the eCRF. Imputed dates for the start date or end date may be used to calculate duration (Section 7.11.1).

## 6.2.2 Clinical Laboratory Variables

Clinical laboratory variables are raw values (i.e., values at each scheduled visit) and changes from baseline for chemistry, hematology and urinalysis parameters at Weeks 2, 4, 8 and Week 10.

SAP Final Version 2.0

## 6.2.3 Vital Signs

Vital signs variables are raw values (i.e., values at each scheduled visit) and changes from baseline in systolic blood pressure (SBP), diastolic blood pressure (DBP) and pulse rate at Day 1 2-hours post dose, Weeks 2, 4, Week 8/EOT and Week 10. Orthostatic SBP, DBP and pulse rate are assessed on Day 1 pre-dose, Day 1 2-hours post dose, Week 8/EOT (triplicate supine measurements approximately 1 minute apart [-3, -2, -1 minutes before standing] followed by a single standing measurement approximately 3 minutes after standing). Single resting measurements of SBP, DBP and pulse rate are measured on at Screening, Weeks 2, 4 and Week 10.

Orthostatic vital signs (SBP, DBP, pulse rate) will be derived for each subject as follows:

| | | 0 |
|---|---|---|
| Analysis Time point | Item | Derivation |
| Baseline, Treatment period | Average supine result | Average of the non-missing supine triplicates taken approximately 1 minute apart (-3, -2, and -1 minutes before standing). |
| Day 1 2-hours post dose,<br>Week 8/EOT | Orthostatic result | Standing result – Average supine result. |
| | | If the result for standing or average supine is not available, then the result will be set to missing. |

**Table 13** Derivation of Orthostatic Vital Signs

## 6.2.4 Electrocardiograms

The 12-lead electrocardiograms (ECG) scheduled assessments will be made at Baseline, Week 8/EOT and Week 10. The results will be recorded as "normal", "abnormal not clinically significant", or "abnormal clinically significant". Electrocardiogram variables are raw values (categorical) at each scheduled visit and changes from baseline (shift from baseline) at Week 8 and Week 10.

## 6.2.5 Columbia Suicide Severity Rating Scale

The Columbia suicide severity rating scale (C-SSRS) is a questionnaire used for suicide assessment. At screening, the "Screening/Baseline" version is to be used to determine eligibility. During all subsequent visits, the "Since last visit" version is used to monitor on-study suicidal ideation and behavior after the initial assessment. Analysis will mainly focus on two aspects: suicidal ideation and suicidal behavior and they will be derived for each subject as follows using the "Since Last visit" version:

**Sponsor:** Astellas Pharma Global Development, Inc. (APGD)

ISN/Protocol 8062-CL-0101

Table 14 Derivation of Columbia Suicide Severity Rating Scale (C-SSRS) Scores

| <b>Analysis Time Point</b> | C-SSRS Item | Derivation |
|---|---|---|
| Baseline | Suicidal ideation | A "yes" answer to any one of the following five questions from suicidal ideation section on the |
| Treatment period | | C-SSRS. |
| Week 2, | | 1. Wish to be dead |
| Week 4, | | 2. Non-specific active suicidal thoughts |
| Week 8, | | 3. Active suicidal ideation with any methods (not |
| EOT, | | plan) without intent to act |
| Overall double-blind | | 4. Active suicidal ideation with some intent to |
| treatment period | | act, without specific plan |
| 1 | | 5. Active suicidal ideation with specific plan and |
| Follow-up period | | intent |
| Week 10 | | |
| Overall follow-up period | | If a subject answer "yes" to more than one suicidal |
| | | ideation question within a visit window as an |
| | | analysis time point (Section 7.11.5.3 Table 30) the |
| | | worst-case response (i.e. the highest) will be used in |
| | | any summaries. |
| | Suicidal behavior | A "yes" answer to any one of the following five |
| | | questions from suicidal behavior section on the |
| | | C-SSRS. |
| | | 6. Preparatory acts or behavior |
| | | 7. Aborted attempt |
| | | 8. Interrupted attempt |
| | | 9. Actual attempt |
| | | 10. Completed suicide |
| | | If a subject answer "yes" to more than one suicidal |
| | | behavior question within a visit window (Section |
| | | 7.11.5.3 Table 30, at an analysis time point the |
| | | worst-case response (i.e. the highest) will be used in |
| | | any summaries. |
| | Suicidal ideation or | A "yes" answer to any one of the above ten suicidal |
| | behavior | ideation or behavior questions on the C-SSRS. |
| | Self-injurious behavior | A "yes" answer to the following question from |
| | without suicidal intent | suicidal behavior section on the C-SSRS: "Has |
| | | subject engaged in Non-Suicidal Self-Injurious |
| | | Behavior?" |

There will be no imputation for missing answers on questions.

## 6.3 Pharmacokinetic Variables

Pharmacokinetic (PK) sampling will occur on Day 1 in the clinic at approximately 1 to 4 hour(s) after dosing and once at Weeks 2, 4 and 8/EOT. PK samples at weeks 2, 4, and 8/EOT should be evenly split between the following 3 sampling windows: before dosing, 1-4 hours post dose and >4 hours post dose. Time of the last dose and time of sample collection will be captured in the electronic Case Report Form (eCRF) during these visits, as well as the date and time of the last meal in relation to that dose will be captured in the eCRF.

Analysis of ASP8062 and any metabolites (if applicable) will be performed using a validated method at a bioanalytical laboratory specified by the Sponsor.

## 6.4 Other Variables

## 6.4.1 Exposure

For each subject, duration of exposure (defined as length of time on 8 weeks of treatment period) will be calculated in days, using the following formula:

 Duration of exposure = Date of last dose of study drug - Date of first dose of study drug +1,

where the <u>date of first dose of study drug</u> and the <u>date of last dose of study drug</u> are defined as the first study drug dosing date and the last study drug dosing date, as captured in the eCRF. Imputed dates for the first or last dose of study drug may be used to calculate exposure (Section 7.11.1).

## 6.4.2 Percent Overall Compliance

Subjects will be instructed to take 2 tablets once per day, one tablet of 25 mg and 1 tablet of 5 mg.

Percent tablet-count compliance is defined as the number of tablets taken divided by the total number of tablets that should have been taken:

Total number of tablets actually received during 8 weeks of treatment period

Total number of tablets planned to receive during 8 weeks of treatment period

x100

#### Where.

- Total number of tablets actually received during 8 weeks of treatment period = total number of tablets dispensed during 8 weeks of treatment period total number of tablets returned during 8 weeks of treatment period.
- Total number of tablets planned to receive during 8 weeks of treatment period = 2 x duration of exposure. Duration of exposure will be calculated as described in Section 6.4.1

Double-blind study drug compliance for the entire double-blind treatment period will be calculated for subjects whose total number of tablets taken and the complete date of the first dose and the last dose of double-blind study drug are known.

#### 6.4.3 Previous and Concomitant Medication

Previous and concomitant non-medication therapy
 A previous non-medication therapy (screening/wash-out) is defined as any non-medication therapy administered up to the last day of screening/washout (i.e., prior to the baseline diary run-in).

A previous non-medication therapy (baseline diary run-in) is defined as any non-medication therapy administered after the last day of screening/washout and before the first dose of double-blind study drug.

**Sponsor:** Astellas Pharma Global Development, Inc. (APGD)

ISN/Protocol 8062-CL-0101

SAP Final Version 2.0

A concomitant non-medication therapy (double-blind treatment period) is defined as any non-medication therapy administered between the first dose (inclusive) of double-blind study drug and the last dose of double-blind study drug (inclusive).

A concomitant non-medication therapy (follow-up period) is defined as any non-medication therapy administered after the last dose of double-blind study drug.

Previous and concomitant medication

A previous medication (screening/wash-out) is defined as any medication taken up to the last day of screening/washout (i.e., prior to the baseline diary run-in).

A previous medication (baseline diary run-in) is defined as any medication taken after the last day of screening/washout and before the first dose of double-blind study drug.

A concomitant medication (double-blind treatment period) is defined as any medication taken between the first dose (inclusive) of double-blind study drug and the last dose of double blind study drug (inclusive).

A concomitant medication (follow-up period) is defined as any medication taken after the last dose day of double-blind study drug.

## 6.4.4 Time Since Onset of Fibromyalgia Symptoms and Time Since Diagnosis

- Time since onset of FM symptoms (years) = (Informed consent date -date FM symptoms started + 1)/365.25
- Time since FM diagnosis (years) = (Informed consent date date of FM diagnosis + 1)/365.25.

Imputed dates for the date FM symptoms started and FM diagnosis may be used to calculate both of these endpoints as described in Section 7.11.1

## 6.4.5 Mini-International Neuropsychiatric Interview

The M.I.N.I. International Neuropsychiatric Interview (M.I.N.I 7.0) is a short, structured diagnostic interview administered by trained personnel. The instrument captures the major Axis I psychiatric disorders in Diagnostic and Statistical Manual of Mental Disorders (DSM-V) and International Statistical Classification of Diseases and Related Health Problems (ICD-10). Each module begins with screening questions that are answered yes or no. A negative response in the screening algorithm advances the interview to the next module, whereas a positive response will prompt additional questions that ask subjects to characterize behavior with "yes" or "no" responses. The final number of YESs or NOs allows the coding a final evaluation per module by Yes/No answer (according to time recall) or severity (according to module): current, in early remission and in remission. The M.I.N.I. 7.0 will be completed at Screening and any diagnosis identified from the M.I.N.I will be captured in the eCRF.

## 6.4.6 Widespread Pain Index and Symptom Severity Scale score

The Widespread Pain Index (WPI) and Symptom Severity (SS) scale score will be completed by the clinician on a tablet device during the Screening visit.

The WPI is a checklist of 19 non-articular body parts classified in 5 body regions. The body parts are checked if pain/tenderness is observed. The WPI global score is the sum of body parts checked as presence of pain and ranges from 0 to 19.

The SS Scale is comprised of two parts:

- First part: evaluation of 3 key-symptoms (fatigue, waking unrefreshed and cognitive symptoms) over the past week. The severity of these symptoms will be measured on a 4-point response scale (from 0 = no problem to 3 = severe).
  - The score for the first part is the sum of the item scores and ranges from 0 to 9.
- Second Part: presence evaluation (1=presence and 0=absence) of 3 other somatic symptoms (headaches, pain/cramps in lower abdomen and depression) during the previous 6 months.

The score for the second part is the sum of the item scores and ranges from 0 to 3.

The SS Scale score is the sum of the first and the second part scores and ranges from 0 to 12.

## 6.4.7 Complex Medical Symptoms Inventory

The Complex Medical Symptoms Inventory (CMSI) is designed to aid clinicians in collecting information from fibromyalgia patients regarding their disease-specific symptoms and to characterize the diagnosis. The inventory contains 2 parts: a symptom checklist to be completed by patients, and a diagnostic inventory completed by the clinician. In this study, only the symptom checklist will be utilized.

The symptom checklist contains 39 items (males) or 41 items (females). For each symptom question, subjects mark a box to indicate if the symptom: 1) has occurred for at least 3 months in the past year, and/or 2) has occurred for a 3-month period during their lifetime. Only the boxes that apply should be checked. The CMSI will be completed on the tablet device by the subject at Baseline Diary Run-In (Visit 2). The CMSI total score is the sum of the number of items that the subject checks as either occurring for at least 3 months in the past year and/or has occurred for a 3-month period during their lifetime. The CMSI total score at baseline will be calculated and ranges from 0 to 39 for males and 0 to 41 for females. Baseline is defined as the last assessment on or prior to the first dose day (Day 1) of double-blind study drug.

## 7 STATISTICAL METHODOLOGY

## 7.1 General Considerations

For continuous variables, descriptive statistics will include the number of subjects (n), mean, standard deviation (SD) and/or standard error (SE), median, minimum and maximum. When needed, the use of other percentiles (e.g. 10%, 25%, 75% and 90%) will be mentioned in the relevant section. Frequencies and percentages will be displayed for categorical data. Percentages by categories will be based on the number of subjects with no missing data, i.e. will add up to 100%.

Summaries based on FAS and PPS (e.g. disposition, baseline and efficacy data) will be presented by planned treatment group, unless specifically stated otherwise. Safety analysis and other summaries based on SAF will be presented by actual treatment received. For summaries which present both absolute values over time and change from baseline values over time the number of subjects used to calculate the descriptive statistics will be those who have non-missing data at each analysis visit and at baseline. For endpoints which include mBOCF, LOCF or mLOCF imputation the descriptive statistics will be calculated after the imputation has been performed.

Unless otherwise specified, statistical comparisons will be made using one-sided tests at the  $\alpha$ =0.05 significance level and two-sided 90% confidence intervals (CIs) will be presented when applicable. When two-sided p-values are presented statistical comparisons will be made using an  $\alpha$ =0.1 significance level.

The pooled site will be used in all statistical models that include the "center" as a factor. The pooling sites algorithm is provided in Section 7.11.6

All data, including observed and derived data, will be presented in subject data listings.

All data processing, summarization, and analyses will be performed using SAS® Version 9.3 or higher on Unix. Specifications for table, figures, and data listing formats can be found in the TLF specifications for this study.



#### **Definition of Study Day:**

The number of study days relative to the first dose date of study drug (Study Day), is calculated as:

- Study Day = Date of assessment Date of first dose of study drug +1, when the date of assessment is <u>on or after</u> the date of first dose of study drug
- Study Day = Date of assessment Date of first dose of study drug, when the date of
  assessment is before the date of first dose of study drug

where the date of first dose of study drug is defined in Section 6.4.1

The day of the first dose of study drug is defined as Study Day 1, while the day before the date of first dose of study drug (i.e., Randomization visit) is defined as Study Day -1 (there is no Study Day 0).

**Sponsor:** Astellas Pharma Global Development, Inc. (APGD)

SAP Final Version 2.0 ISN/Protocol 8062-CL-0101

For daily average pain scores assessed by NRS any data captured in the e-diary up to 2am in the morning of the following day will be assigned to the previous day in the derivation of Study Day.

## **Definition of Follow-up Day:**

The number of study days relative to the last dose date of study drug (Follow-up Day), is calculated as:

Follow-up Day = Date of assessment – Date of last dose of study drug where the date of last dose of study drug up is defined in Section 6.4.1

Follow-up Day will equal zero on the day of the last dose of study drug and positive values will indicate days during the follow-up period.

For daily average pain scores assessed by NRS any data captured in the ediary up to 2 am in the morning of the following day will be assigned to the previous day in the derivation of Follow-up Day.

## **Definition of Treatment Period:**

Time from Study Day 1, through to Follow-up Day 4.

#### **Definition of Efficacy Follow-up Period:**

Time from Follow-up Day 5 through to Follow-up Day 28.

## **Definition of Safety Follow-up Period:**

Time from Follow-up Day 5 through to Follow-up Day 30.

#### 7.2 **Study Population**

#### 7.2.1 **Disposition of Subjects**

The following subject data will be presented:

- Number of subjects with informed consent, discontinued during screening/wash-out, entered the baseline diary run-in, discontinued prior to randomization, randomized for all subjects with informed consent ('Total' overall only);
- Number and percentage of subjects who were randomized, took study drug, did not take study drug, in the analysis sets by treatment group and 'Total' over all treatment groups for all randomized subjects;
- Number and percentage of subjects who completed and discontinued the screening/washout, and primary reason for discontinuing screening/wash-out for all subjects with informed consent ('Total' overall only);
- Number and percentage of subjects who completed and discontinued prior to randomization, and primary reason for discontinuing prior to randomization for all subjects who came for randomization visit ('Total' overall only);

 Number and percentage of subjects who completed and discontinued treatment, and primary reason for treatment discontinuation by treatment group and 'Total' over all treatment groups for all randomized subjects, SAF and FAS;

- Number and percentage of subjects completed and discontinued the follow-up period, and primary reason for discontinuing the follow-up period by treatment group and 'Total' over all treatment groups for all randomized subjects and SAF;
- Number and percentage of subjects who completed and discontinued treatment at each visit, by primary reason for treatment discontinuation by treatment group and 'Total' over all treatment groups for all randomized subjects, SAF and FAS;
- Number and percentage of subjects excluded from PPS by reason for exclusion defined in Section 5.2.1 by treatment group and 'Total' over all treatment groups for FAS; and
- Number and percentage of subjects for each protocol version by treatment group and 'Total' over all treatment groups for randomized subjects, as well as, number and percentage of subjects for each protocol version for screen failures (subjects who discontinued during screening/wash-out, or prior to randomization) and Total Number of subjects enrolled (i.e. including Screen Failures).

A stacked bar plot of cumulative discontinuation rates (colored by primary reason for discontinuation) overall and at each visit by treatment group will be produced for the SAF.

#### 7.2.2 Protocol Deviations

Protocol deviations as defined in the study protocol (Section 8.1.6 Protocol Deviations) will be assessed for all randomized subjects. The number and percentage of subjects meeting any criteria will be summarized for each criterion and overall, by treatment group and total as well as by study site. Subjects deviating from a criterion more than once will be counted once for the corresponding criterion. Any subjects who have more than one protocol deviation will be counted once in the overall summary. A data listing will be provided by site and subject.

The protocol deviation criteria will be uniquely identified in the summary table and listing. The unique identifiers will be as follows:

- PD1 Entered into the study even though they did not satisfy entry criteria,
- PD2 Developed withdrawal criteria during the study and was not withdrawn,
- PD3 Received wrong treatment or incorrect dose,
- PD4 Received excluded concomitant treatment.

#### 7.2.3 Demographic and Other Baseline Characteristics

No hypothesis testing will be performed comparing treatment groups for demographic and other baseline characteristics.

## 7.2.3.1 Demographics

Demographic characteristics will be summarized by descriptive statistics for the following variables listed in Table 15 This will be done for all randomized subjects, as well as for the SAF, FAS and PPS by treatment group and 'Total' over all treatment groups.

**Table 15 Demographic Characteristics** 

| Characteristic | Summarized as | Categories |
|---|---|---|
| Age (years) | Continuous | |
| Weight (kg) | Continuous | |
| Height (cm) | Continuous | |
| BMI (kg/m <sup>2</sup> ) | Continuous | |
| Sex | Categorical | <ul><li>Male</li><li>Female</li><li>Unknown</li></ul> |
| Race | Categorical | <ul> <li>White</li> <li>Black or African American</li> <li>Asian</li> <li>American Indian or Alaska Native</li> <li>Native Hawaiian or Other Pacific Islander</li> <li>Other</li> </ul> |
| Ethnicity | Categorical | <ul><li>Not Hispanic or Latino</li><li>Hispanic or Latino</li></ul> |
| Age group | Categorical | <ul> <li>&lt; 45 years</li> <li>≥ 45 to &lt; 65 years</li> <li>≥ 65 years</li> </ul> |
| EudraCT Age group | Categorical | <ul> <li>≥ 18 to ≤ 64 years</li> <li>≥ 65 to ≤ 84 years</li> </ul> |
| BMI group 1 | Categorical | • $< 25 \text{ kg/m}^2$<br>• $≥ 25 \text{ to} < 30 \text{ kg/m}^2$<br>• $≥ 30 \text{ kg/m}^2$ |
| BMI group 2 | Categorical | $ \begin{array}{l} \bullet & < 30 \text{ kg/m}^2 \\ \bullet & \geq 30 \text{ kg/m}^2 \end{array} $ |

Number and percentage of subjects randomized in each site will be presented by treatment group and 'Total' over all treatment groups for randomized subjects. In addition, number and percentage of pooled sites and the combination of sites into pooled sites will be summarized by treatment group and overall for the FAS.

## 7.2.3.2 Fibromyalgia and Targeted Medical History

Fibromyalgia and targeted medical history will be summarized by descriptive statistics for the following variables listed in Table 16 This will be done for all randomized subjects, the SAF, FAS and PPS by treatment group and 'Total' over all treatment groups.

 $\textbf{Sponsor:} \ Astellas \ Pharma \ Global \ Development, \ Inc. \ (APGD)$ 

ISN/Protocol 8062-CL-0101

 Table 16
 Fibromyalgia Diagnosis and Targeted Medical History

| Characteristic | Summarized as | Categories |
|---|---|---|
| Time since FM diagnosis (years) | Continuous | |
| Time since onset of FM symptoms (years) | Continuous | |
| Currently treated for FM | Categorical | <ul><li>Yes</li><li>No</li></ul> |
| History of Major Depressive Disorder (MDD) as assessed by M.I.N.I. | Categorical | <ul><li>No</li><li>Yes</li><li>No</li></ul> |
| Ongoing MDD (only for subjects with a History of MDD) | Categorical | <ul><li>Yes</li><li>No</li></ul> |
| Currently Treated with Medication for MDD (only for subjects with a History of MDD) | | <ul><li>Yes</li><li>No</li></ul> |
| HADS Depression total score | Continuous | |
| HADS Depression group | Categorical | <ul> <li>Normal (0 to 7)</li> <li>Mild mood disturbance (8 to 10)</li> <li>Moderate mood disturbance (11 to 14)</li> <li>Severe mood disturbance (15 to 21)</li> </ul> |
| C-SSRS Item: | Categorical | For each item: • Yes • No |
| History of Temporomandibular<br>Disorders | Categorical | <ul><li>Yes</li><li>No</li></ul> |
| History of Irritable Bowel Syndrome | Categorical | <ul><li>Yes</li><li>No</li></ul> |
| History of Chronic Tension Type<br>Headache | Categorical | <ul><li>Yes</li><li>No</li></ul> |
| History of Migraine | Categorical | <ul><li>Yes</li><li>No</li></ul> |
| History of Chronic Low Back Pain | Categorical | <ul><li>Yes</li><li>No</li></ul> |
| History of Myalgic<br>Encephalomyelitis/Chronic Fatigue<br>Syndrome | Categorical | <ul><li>Yes</li><li>No</li></ul> |
| Table continued on next page | | |

| Characteristic | Summarized as | Categories |
|---|---|---|
| History of Interstitial Cystitis/Painful | Categorical | • Yes |
| Bladder Syndrome | | • No |
| History of Endometriosis (Females | Categorical | • Yes |
| Only) | | • No |
| History of Vulvodynia (Females | Categorical | • Yes |
| Only) | | • No |
| Alcohol History | Categorical | • Never |
| | | <ul> <li>Current</li> </ul> |
| | | • Former |
| History of Alcohol Use Disorder | Categorical | • Yes |
| (only for subjects with current or | | • No |
| former Alcohol History) | | |
| History of Drug Use | Categorical | • Never |
| | | <ul> <li>Current</li> </ul> |
| | | • Former |
| History of Substance Use Disorder | Categorical | • Yes |
| (only for subjects with current or | | • No |
| former History of Drug Use) | | |
| First or Second Degree Family | Categorical | For each Family History: |
| History of | | • Yes |
| <ul> <li>Fibromyalgia</li> </ul> | | • No |
| <ul> <li>Depression</li> </ul> | | |
| <ul> <li>Bipolar disorder</li> </ul> | | |

CMSI: Complex Medical Symptom Inventory, C-SSRS: Columbia Suicide Severity Rating Scale, FM: Fibromyalgia, HADS: Hospital Anxiety and Depression Scale, MDD: Major Depressive Disorder, M.I.N.I: Mini-International Neuropsychiatric Interview,

## 7.2.3.3 Fibromyalgia Related Baseline Disease Characteristics

Fibromyalgia related baseline disease characteristics will be summarized by descriptive statistics for the following variables listed in Table 17 This will be done for all randomized subjects, the SAF, FAS and PPS by treatment group and 'Total' over all treatment groups.

 Table 17
 Fibromyalgia Related Baseline Disease Characteristics

| Characteristic | Summarized as | Categories |
|---|---|---|
| Baseline mean daily average pain score assessed by NRS | Continuous | |
| Baseline mean daily average pain score assessed by NRS group | Categorical | <ul> <li>No pain: 0</li> <li>Mild: &gt; 0 to &lt; 4</li> <li>Moderate: ≥ 4 to &lt; 7</li> <li>Severe: ≥ 7 to 10</li> </ul> |
| WPI | Continuous | |
| SS scale score | Continuous | |
| Tender point count | Continuous | |
| PGIS | Categorical | <ul> <li>No symptoms</li> <li>Very mild</li> <li>Mild</li> <li>Moderate</li> <li>Severe</li> <li>Very severe</li> </ul> |
| Table continued on next page | · | |



CMSI: Complex Medical Symptom Inventory, FIQR: Fibromyalgia Impact Questionnaire Revised, FM: Fibromyalgia;

NRS: Numerical Rating Scale; PGIS: Patient Global Impression of Severity, SS: Symptom severity, WPI: Widespread pain index.

## 7.2.3.4 Medical History

Medical history is coded in Medical Dictionary for Regulatory Activities (MedDRA), and will be summarized by System Organ Class (SOC) and Preferred Term (PT) as well as by PT alone, by treatment group and "Total" over all treatment groups for the SAF.

<sup>\*</sup> CMSI will be split into three groups using the CMSI total score at baseline: more centrally driven FM pain (≤ 1st tertile); non-specific FM pain (> 1st tertile to < 3rd tertile) and more peripherally driven FM pain (≥ 3rd tertile);

## 7.2.4 Previous and Concomitant Medications

The following will be presented using the SAF:

- All previous medications prior to the baseline diary run-in
- All previous medications taken for any pain (i.e., FM pain only or FM pain and Other type of pain or Other type of pain only) prior to baseline diary run-in,
- All previous medications taken for FM pain (FM pain only or FM pain and Other type of pain) prior to baseline diary run-in,

SAP Final Version 2.0

- All previous medications during baseline diary run-in,
- All previous medications taken for any pain during baseline diary run-in,
- All previous medications taken for FM pain during baseline diary run-in,
- All concomitant medications during the double-blind treatment period,
- All concomitant medications taken for any pain during the double-blind treatment period,
- All concomitant medications taken for FM pain during the double-blind treatment period,
- All concomitant medications taken during the follow-up period,
- All concomitant medications taken for any pain during the follow-up period, and
- All concomitant medications taken for FM pain during the follow-up period.

Previous and concomitant medications are coded with World Health Organization Drug Dictionary (WHO-DD). Each of the above will be summarized by therapeutic subgroup (ATC 2nd level) and chemical subgroup (ATC 4th level) and preferred WHO name by treatment group and 'Total' over all treatment groups. Subjects taking the same medication multiple times will be counted once per medication and investigational period. A medication which can be classified into several chemical and/or therapeutic subgroups is presented in all chemical and therapeutic subgroups. All previous medications taken for any pain during baseline diary runin; all concomitant medications taken for any pain during the double blind treatment period and all concomitant medications taken for any pain during the follow-up period will also be summarized by preferred WHO name by treatment group and 'Total' over all treatment groups.

In addition to the above summaries an overview of previous medications taken prior to the baseline diary run-in and previous medications during the baseline diary run-in taken to treat pain, will be produced. This will summarize the number and percentage of subjects in each of the following categories for each treatment group and 'Total' over all treatment groups:

- Any pain (i.e. FM pain only; or FM pain and Other type of pain; or Other type of pain only),
- FM pain (i.e. FM pain only; or FM pain and Other type of pain),
- FM pain only,
- FM pain and Other type of pain,

As with previous medication, concomitant medication (double-blind treatment period) and concomitant medication (follow-up period) taken to treat pain will be summarized for each treatment group and 'Total' over all treatment groups for the above categories.

The listing will only contain data of the subjects who actually used previous and concomitant medications.

## 7.2.5 Previous and Concomitant Non-Medication Therapy

The following will be presented using the SAF:

- All previous non-medication therapies prior to baseline diary run-in,
- All previous non-medication therapies received for any pain (i.e., FM pain only or FM pain and Other type of pain or Other type of pain only) prior to baseline diary run-in,
- All previous non-medication therapies received for FM pain (FM pain only or FM pain and Other type of pain) prior to baseline diary run-in,
- All previous non-medication therapies received during baseline diary run-in,
- All previous non-medication therapies received for any pain during baseline diary run-in,
- All previous non-medication therapies received for FM pain during baseline diary run-in,
- All concomitant non-medication therapies received during the double-blind treatment period,
- All concomitant non-medication therapies received for any pain during the double-blind treatment period,
- All concomitant non-medication therapies received for FM pain during the double-blind treatment period,
- All concomitant non-medication therapies received during the follow-up period,
- All concomitant non-medication therapies received for any pain during the follow-up period, and
- All concomitant non-medication therapies received for FM pain during the follow-up period.

Each of the above will be summarized by treatment group and 'Total' over all treatment groups for:

- Normal Daily Exercise Routines,
- Chiropractic Care,
- Physical Therapy,
- Psychotherapy,
- Massage therapy, and
- Other.

Subjects receiving the same non-medication therapy multiple times will be counted once per medication and investigational period.

In addition to the above summaries an overview of previous non-medication therapies prior to the baseline diary run-in and previous non-medication therapies during the baseline diary run-in received to treat pain, the number and percentage of subjects with the following

categories will be summarized for each treatment group and 'Total' over all treatment groups:

- Any pain (i.e. FM pain only; or FM pain and Other type of pain; or Other type of pain only),
- FM pain (i.e. FM pain only; or FM pain and Other type of pain),
- FM pain only,
- FM pain and Other type of pain,

As with previous non-medication therapy, concomitant non-medication therapy (double-blind treatment period) and concomitant non-medication therapy (follow-up period) will be summarized for each treatment group and 'Total' over all treatment groups for the above categories.

The listing will only contain data of the subjects who actually used previous and concomitant non-medication therapies.

## 7.3 Study Drugs

## 7.3.1 Exposure

Duration of exposure will be summarized by treatment group and 'Total' over all treatment groups in three ways for the SAF:

- Descriptive statistics will be presented for the total number of days a subject was exposed to study drug.
- Number and percentage of subjects in each of the following mutually exclusive extent of exposure categories:
  - o 1 to 7 days,
  - o 8 to 14 days,
  - o 15 to 28 days,
  - o 29 to 48 days,
  - o 49 to 64 days,
  - $\circ \geq 65 \text{ days}$
- Number and percentage of subjects in the following cumulative extent of exposure time categories:
  - $\circ \geq 1 \text{ day},$
  - $\circ \geq 8 \text{ days};$
  - $\circ \geq 15 \text{ days}$
  - $\circ \geq 29$  days,
  - $\circ \geq 49 \text{ days}$
  - $\circ \geq 65$  days.

## 7.3.2 Treatment Compliance

Overall compliance with the dosing schedule will be examined for subjects in the SAF whose total study drug count and first and last days of treatment are known.

Percent overall compliance will be summarized by treatment group and 'Total' over all treatment groups in two ways for the SAF:

- Descriptive statistics for percent overall compliance.
- Number and percentage of subjects in the following categories of percent overall compliance:
  - $\circ$  < 50%,
  - $\circ > 50\%$  to < 80%,
  - $\circ > 80\%$  to < 100%,
  - $\circ = 100\%$
  - $\circ > 100\%$  to < 120%,
  - $\circ \geq 120\%$ .

## 7.4 Analysis of Efficacy

Efficacy analyses will be performed using the FAS and the PPS where indicated. No formal hypothesis testing of comparison between treatment groups will be performed for the efficacy data during the follow-up period i.e., descriptive statistics will be used to summarize the continuous efficacy variables and frequencies and percentages will be used to summarize the categorical efficacy data.

## 7.4.1 Analysis of Primary Endpoint(s)

Analysis of the primary efficacy endpoint will be performed on the FAS and the PPS. Table 18 describes the primary analysis and sensitivity analyses that will be performed for the primary efficacy endpoint.

Table 18 Summary of the Primary and Sensitivity Analyses for the Primary Efficacy Endpoint

| Variable | Imputation | Analysis Set | Analysis Type |
|---|---|---|---|
| Change from baseline to Week 8 in mean daily average pain score assessed by NRS (Primary Analysis) | None | FAS | MMRM analysis of change from baseline <sup>a</sup> |
| Change from baseline to Week 8 in mean daily average pain score assessed by NRS (Sensitivity Analysis) | Discontinuation-<br>reason based<br>multiple imputation <sup>b</sup> | FAS | MMRM analysis of change from baseline <sup>a</sup> |
| Change from baseline to Week 8 in mean daily average pain score assessed by NRS (Sensitivity Analysis) | mBOCF <sup>c</sup> | FAS | ANCOVA analysis of change from baseline |
| Change from baseline to Week 8 in mean daily average pain score assessed by NRS (Sensitivity Analysis) | None | PPS | MMRM analysis of change from baseline <sup>a</sup> |

<sup>&</sup>lt;sup>a</sup>MMRM analysis uses data from baseline and change from baseline data at Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7 and Week 8 time points.

<sup>&</sup>lt;sup>b</sup>Discontinuation-reason based multiple imputation (MI) will use a "Jump to Reference" algorithm (where placebo is the reference group) for subjects who discontinue due to lack of efficacy or AEs and standard regression-based MI for subjects with missing data for other reasons.

<sup>&</sup>lt;sup>c</sup>mBOCF is defined as imputation by baseline observation carried forward for subjects who discontinue due to lack of efficacy or AEs, and imputation by last observation carried forward for subjects with missing data at Week 8 for other reasons.

SAP Final Version 2.0

ISN/Protocol 8062-CL-0101

## 7.4.1.1 Primary Analysis of Primary Endpoint

The hypothesis for comparison of mean change from baseline between ASP8062 and placebo is shown below:

 $H_0$ : The mean change from baseline to Week 8 in mean daily average pain score assessed by NRS (0 to 10 scale) for ASP8062 30 mg once daily group is same as (or higher, i.e., worse than) the placebo group.

**H**<sub>1</sub>: The mean change from baseline to Week 8 in mean daily average pain score assessed by NRS (0 to 10 scale) for ASP8062 30 mg once daily group is less than the placebo group.

The change from baseline in mean daily average pain score to Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7 and Week 8 will be analyzed using a mixed-effect, repeated measures (MMRM) model including treatment, center (pooled where necessary), time (study Week 1 to 8), and treatment-by-time interaction as fixed effects, baseline mean daily average pain score and baseline mean daily average pain score-by-time interaction as covariates. The treatment group contrasts for change from baseline to Week 8 will be the primary statistical inference obtained from this model.

This analysis will utilize observed data, and there will be no imputation for missing data. Parameters will be estimated using restricted maximum-likelihood and the Kenward-Roger approximation will be used to estimate denominator degrees of freedom and adjust SEs.

An unstructured variance-covariance structure will be used to model the within-subject errors. If the fit of the unstructured covariance structure fails to converge, the following covariance structures will be tried in order until convergence is reached: heterogeneous Toeplitz (for efficacy endpoints captured in e-diary only, i.e. mean daily average pain score assessed by NRS followed by compound symmetry.

Residual plots of scaled residuals will be used to check the fit of the model and assess whether there is any evidence of non-normality.

From the MMRM model the following results will be presented:

- Least squares (LS) mean estimates, SE and 2-sided 90% confidence interval (CI) for mean change from baseline to each analysis time-point (Week 1 to Week 8) within a treatment group (ASP8062, placebo),
- The difference in LS means for ASP8062 versus placebo, SE for the difference and 2-sided 90% CI for the difference at each analysis time-point,
- One-sided p-value for ASP8062 versus placebo at each analysis time-point, and
- Two-sided p-value for treatment-by time interaction.

An overlay plot will be provided for LS mean change from baseline from the MMRM analysis and mean change from baseline from the follow-up period +/- SE vs analysis time-point by treatment group.

## 7.4.1.2 Sensitivity Analyses of Primary Endpoint

The following sensitivity analyses will be performed for the primary efficacy endpoint to assess the robustness of the primary analysis.

## Discontinuation-reason based multiple imputation

The MMRM analysis that will be used to perform the primary analysis of the primary endpoint assumes that missingness is at random. That is, the model assumes that the trajectory of mean daily average pain scores over time for subjects who withdraw is similar to the trajectory for those observed in their own treatment arm which is valid so long as that assumption is reasonable.

Discontinuation-reason based multiple imputation (MI) will be used to examine the sensitivity of the primary analysis results to departures from that underlying assumption and will assess a situation where data for subjects who discontinue early follow a pattern which is missing not at random. Specifically, MI will be used for imputation of any missing data, using "Jump to Reference" algorithm (where placebo is the reference group) [Carpenter et al. 2013] for subjects who discontinue due to lack of efficacy or AEs and standard regression-based MI for subjects with missing data for other reasons. The analysis will be implemented using the general three-step process (imputation phase, followed by analysis phase, followed by pooling phase) described in O'Kelly and Ratitch, 2014.

- 1. The imputation phase will implement MI via sequential modelling for both the "Jump to Reference" algorithm and standard regression-based MI. In particular, when implementing the "Jump to Reference" algorithm via sequential modelling, this means that only baseline values are used in the imputation of missing values for subjects in the ASP8062 30 mg once daily group who discontinue due to lack of efficacy or AEs (this variation of the "Jump to Reference" algorithm is also referred to as the "Unconditional Reference" approach). The imputation phase will generate *M* imputed datasets, where *M*=100.
- 2. The analysis phase will perform the primary MMRM analysis model of the primary efficacy endpoint as described in Section 7.4.1.1 for each of the M=100 imputed datasets (which now contain complete data, where missing data have been filled in).
- 3. Rubin's rules will be used to generate an overall set of pooled results which combines the analysis results from the M=100 imputed datasets.

The overall set of pooled results will present:

- Least squares (LS) mean estimates, SE and 2-sided 90% confidence interval (CI) for mean change from baseline to Week 8 within a treatment group (ASP8062, placebo),
- The difference in LS means for ASP8062 versus placebo, SE for the difference and 2-sided 90% CI for the difference at Week 8,
- One-sided p-value for ASP8062 versus placebo at Week 8, obtained using the difference in the LS means.
- Descriptive summary statistics at Week 8 will be derived using the mean of the M=100 imputed datasets.

Descriptive summaries and plots will be used to explore the pattern of missingness are described in Section 7.2.1

#### Modified baseline observation carried forward

Prior to any analysis mBOCF will be used to impute any missing Week 8 data. Modified baseline observation carried forward is defined as imputation by BOCF for subjects who discontinue due to lack of efficacy or AEs, and imputation by LOCF for subjects with missing data at Week 8 for other reasons. The imputed change from baseline to Week 8 data will be analyzed using ANCOVA with treatment group and center (pooled site) as fixed effects and baseline value as a covariate.

The ANCOVA will present LS mean estimates, SE for the LS means and two-sided 90% CI for change from baseline to Week 8 within a treatment group (ASP8062, placebo). For comparisons between ASP8062 and placebo for the change from baseline to Week 8, the ANCOVA model will present the difference in LS mean estimates, SE and corresponding 2-sided 90% CI. The differences in LS mean estimates will be used to obtain 1-sided p-values for ASP8062 versus placebo.

#### Per-protocol analysis

The same analysis of the primary efficacy endpoint as described in Section 7.4.1.1 will be repeated using the PPS.

## 7.4.1.3 Subgroup analysis

The subgroup analysis of the primary efficacy endpoint is described in Section 7.8.1

## 7.4.2 Analysis of Secondary Endpoints

Analysis of secondary efficacy endpoints will be performed on the FAS. Analyses of select secondary endpoints will be performed on the PPS as specified in Table 19

Table 19 Summary of the Analyses for the Secondary Efficacy Variables

| Variable | Imputation | Analysis<br>Set | Analysis Type |
|---|---|---|---|
| Percentage of subjects achieving ≥ 30% (or ≥ 50%) reduction from baseline to Week 8 in mean daily average pain score assessed by NRS where all subjects with missing Week 8 data are classified as non-responders | BOCF | FAS | Fisher's exact test |
| Percentage of subjects achieving $\geq$ 30% (or $\geq$ 50%) reduction from baseline to Week 8 in mean daily average pain score assessed by NRS (Sensitivity analysis) | mBOCF <sup>c</sup> | FAS | Fisher's exact test |
| Percentage of subjects achieving $\geq$ 30% (or $\geq$ 50%) reduction from baseline to Week 8 in mean daily average pain score assessed by NRS where all subjects with missing Week 8 data are classified as non-responders (Sensitivity analysis) | BOCF | PPS | Fisher's exact test |
| Table continued on next page | | | |

| Variable | Imputation | Analysis<br>Set | Analysis Type |
|---|---|---|---|
| Percentage of subjects achieving $\geq 30\%$ (or $\geq 50\%$ ) reduction from baseline to EOT in mean daily average pain score assessed by NRS | LOCF | FAS | Fisher's exact test |
| Change from baseline to Week 2, Week 4 and Week 8 for the FIQR function, symptoms and overall impact subscales | None | FAS | MMRM analysis of change from baseline <sup>a</sup> |
| Change from baseline to Week 8 for the FIQR function, symptoms and overall impact subscales (Sensitivity analysis) | Discontinuation-<br>reason based<br>multiple<br>imputation <sup>b</sup> | FAS | MMRM analysis of change from baseline <sup>a</sup> |
| Change from baseline to Week 8 for the FIQR function, symptoms and overall impact subscales (Sensitivity analysis) | None | PPS | MMRM analysis of change from baseline <sup>a</sup> |
| Change from baseline to Week 8 for the FIQR function, symptoms and overall impact subscales (Sensitivity Analysis) | mBOCF <sup>c</sup> | FAS | ANCOVA analysis of change from baseline |
| Change from baseline to EOT for the FIQR function, symptoms and overall subscales | LOCF | FAS | ANCOVA analysis of change from baseline |
| Overall subject improvement assessed by PGIC at Week 2, Week 4 and Week 8 | mBOCF <sup>c</sup> | FAS | Proportional odds model |
| Overall subject improvement assessed by PGIC at Week 2 and Week 4 (Sensitivity analysis) | LOCF | FAS | Proportional odds model |
| Overall subject improvement assessed by PGIC at EOT | LOCF | FAS | Proportional odds model |

<sup>&</sup>lt;sup>a</sup>MMRM analysis uses data from baseline and change from baseline data at Week 2, Week 4 and Week 8 time points.

The following secondary binary response endpoints (responder, non-responder; as defined in Section 6.1.2) will be analyzed using the Fisher's exact test for ASP8062 versus placebo:

- Percentage of subjects achieving ≥ 30% (or ≥ 50%) reduction from baseline to Week 8 in mean daily average pain score assessed by NRS where all subjects with missing Week 8 data are classified as non-responders,
- Percentage of subjects achieving ≥ 30% (or ≥ 50%) reduction from baseline to Week 8 in mean daily average pain score assessed by NRS where mBOCF is used to impute a responder status for subjects with missing Week 8 data, and
- Percentage of subjects achieving ≥ 30% (or ≥ 50%) reduction from baseline to EOT in mean daily average pain score assessed by NRS.

Summary statistics will show the number and percentage of subjects who show response for each treatment group, 2-sided 90% CI for the percentage within each treatment group (ASP8062, placebo) calculated using the exact unconditional approach, difference in

<sup>&</sup>lt;sup>b</sup>Discontinuation-reason based multiple imputation (MI) will use a "Jump to Reference" algorithm (where placebo is the reference group) for subjects who discontinue due to lack of efficacy or AEs and standard regression-based MI for subjects with missing data for other reasons.

<sup>&</sup>lt;sup>c</sup>mBOCF is defined as imputation by baseline observation carried forward for subjects who discontinue due to lack of efficacy or AEs, and imputation by LOCF for subjects with missing data at the specific analysis time point for other reasons.

percentages, 2-sided 90% CI for ASP8062 versus placebo calculated using the exact unconditional approach, and 1-sided p-value. In addition, the above responder analysis will be repeated in the PPS as a sensitivity analysis of the percentage of subjects achieving  $\geq 30\%$  (or  $\geq 50\%$ ) reduction from baseline to Week 8 in mean daily average pain score assessed by NRS where all subjects with missing Week 8 data are classified as non-responders.

The following secondary endpoints will be analyzed using the MMRM analysis as described in Section 7.4.1.1 for the primary efficacy analysis (however with only analysis time-points Week 2, Week 4 and Week 8 included):

• Change from baseline to Week 2, Week 4 and Week 8 for the FIQR function, symptoms and overall impact subscales (where no explicit imputation is performed).

For each endpoint, standard summaries of the MMRM analysis results will be provided, as described in Section 7.4.1.1 This will include an overlay plot. In addition, the MMRM analysis will be repeated in the PPS and also in the FAS under the assumption that data is MNAR using decision-reason based multiple imputation as sensitivity analyses of the change from baseline to Week 8 for the FIQR function, symptoms and overall impact subscales.

The following secondary endpoints will be analyzed using ANCOVA, as described in Section 7.4.1.2 for the second sensitivity analysis of the primary endpoint:

- Change from baseline to Week 8 in FIQR function, symptoms and overall impact subscale scores where mBOCF is used for imputation of missing data at Week 8.
   Modified baseline observation carried forward is defined as imputation by BOCF for subjects who discontinue due to lack of efficacy or AEs, and imputation by LOCF for subjects with missing data at Week 8 for other reasons.
- Change from baseline to EOT in FIQR function, symptoms, and overall impact subscale scores.

For each endpoint, standard summaries of the ANCOVA results, as described in Section 7.4.1.2, will be provided.

The following secondary endpoints will be analyzed using a proportional odds model for ordinal data including treatment group as a factor:

- Overall subject improvement assessed by PGIC at Week 2, Week 4 and Week 8 where mBOCF will be used for subjects with missing data,
- Overall subject improvement assessed by PGIC at Week 2 and Week 4 where LOCF will be used for subjects with missing data, and
- Overall subject improvement assessed by PGIC at EOT.

At each time point, the proportion of subjects in each treatment group achieving each level of response (1 = "Very Much Improved", 2 = "Much improved", 3 = "Minimally Improved", 4 = "No Change", 5 = "Minimally Worse", 6 = "Much Worse", 7 = "Very Much Worse"), will be presented, together with the odds ratio, associated 90% CI based on profile likelihood and 2-sided p-value based on likelihood ratio test for ASP8062 vs placebo. The cumulative logit link will be used to specify the proportional odds model in SAS.















#### 7.4.4 Analysis of Other Variables

Not applicable.

## 7.5 Analysis of Safety

All analysis of safety will be presented by treatment group for SAF, unless specified otherwise. No hypothesis testing will be performed comparing treatment groups for any safety parameters.

#### 7.5.1 Adverse Events

Summaries and listings of serious adverse events (SAEs) and serious TEAEs include SAEs upgraded by the sponsor based on review of the Sponsor's list of Always Serious terms if any upgrade was done.

Duration of AE will be included in all listings and is calculated as described in Section 6.2.1

The coding dictionary for this study will be MedDRA version 20.0. It will be used to summarize AEs by SOC and PT. Standardized MedDRA query (SMQs) will also be used to identify AEs of interest as described in Section 7.5.2

#### 7.5.1.1 Adverse Events Prior to First Dose

The number and percentage of subjects with AEs prior to first dose, as classified by SOC and PT will be summarized for each treatment group.

## 7.5.1.2 Treatment Emergent Adverse Events

An overview table will include the following details:

- Number of TEAEs,
- Number and percentage of subjects with TEAEs,
- Number of drug related TEAEs,
- Number and percentage of subjects with drug related TEAEs,
- Number of serious TEAEs,
- Number and percentage of subjects with serious TEAEs,
- Number of drug related serious TEAEs,
- Number and percentage of subjects with drug related serious TEAEs,
- Number of TEAEs leading to permanent discontinuation of study drug,
- Number and percentage of subjects with TEAEs leading to permanent discontinuation of study drug,

- Number of deaths,
- Number of drug abuse related TEAEs, and
- Number of drug withdrawal related TEAEs.

The above summary will be repeated for TEAEs (treatment period) and TEAEs (follow-up period).

## 7.5.1.3 Treatment Emergent Adverse Events by SOC and/or PT

The number and percentage of subjects with TEAEs, as classified by SOC and PT will be summarized for each treatment group. Summaries will be provided for:

- TEAEs
- TEAEs (treatment period) and TEAEs (follow-up period),
- Drug related TEAEs,
- Serious TEAEs (including number of events),
- Drug related serious TEAEs (including number of events),
- TEAEs leading to permanent discontinuation of study drug,
- Drug related TEAEs leading to permanent discontinuation of study drug,
- TEAEs leading to death (including number of events)
- Drug related TEAEs leading to death (including number of events),
- TEAEs excluding serious adverse events that equal to or exceed a threshold of 5% in any treatment group.

The number and percentage of subjects with TEAEs, as classified by PT only, will be summarized for each treatment group in decreasing order of frequency within the ASP8062 treatment group.

The number and percentage of subjects with TEAEs (including number of events), as classified by SOC and PT will also be summarized by severity to study drug. In the subject count, if a subject has multiple TEAEs with the same SOC or PT, but with differing severity, then the subject will be counted only once with the worst severity. If any of the severity values are missing then the subject will be counted only once with worst severity, i.e. severe. In the adverse event count, the adverse events will be presented in each category they were classified to.

Drug related TEAEs will be presented in a similar way by severity only. When assessing severity for drug-related TEAEs as reported by the investigator, only drug-related TEAEs will be used in the analysis and the worst grade for severity will be chosen as described above.

#### 7.5.2 Adverse Events of Interest

The number and percent of subjects who have a TEAE within the Drug abuse, dependence and withdrawal SMQ (MedDRA 20.0) will be summarized by treatment group.

#### **Drug abuse related TEAEs**

The number and percent of subjects who have a TEAE within the Drug abuse and dependence SMQ (MedDRA 20.0) during the treatment period and follow-up period, as classified by SOC and PT will be summarized by treatment group.

In addition, the number and percent of subjects who have Drug abuse related TEAEs during the treatment period and follow-up period, as defined in Section 10.1 Appendix 1: Drug Abuse Related Adverse Events as classified by PT and lowest level term will be summarized by treatment group.

#### **Drug withdrawal related TEAEs**

The number and percent of subjects who have a TEAE within the Drug withdrawal SMQ (MedDRA 20.0) during the treatment period and follow-up period, as classified by SOC and PT will be summarized treatment group.

In addition, the number and percent of subjects who have withdrawal related TEAEs during the treatment period and follow-up period, as defined in Section 10.2 Appendix 2: Drug Withdrawal Related Adverse Events as classified by SOC and PT will be summarized by treatment group.

## 7.5.3 Clinical Laboratory Evaluation

The baseline visit is the last measurement taken prior to first dose of study drug.

Quantitative clinical laboratory variables, i.e., hematology & coagulation, and biochemistry will be summarized using mean, SD, minimum, maximum and median for each treatment group at each visit. Additionally, a within-subject change will be calculated as the post-baseline measurement minus the baseline measurement and summarized in the same way. Each laboratory result will be classified as low (L), normal (N), or high (H) at each visit according to the laboratory supplied reference ranges.

The number and percentage of subjects below and above the reference range will be summarized for each treatment group at each visit.

For hematology and biochemistry, two types of shift tables will be presented for each treatment group:

- Shift tables of reference range changes from baseline to post-baseline value at each specified time point (low, normal, high), and
- Summary shifts of reference range changes from baseline to post-baseline value at each specified time point (shift from normal or high to low, shift from normal or low to high, categorized increase [shift from low to normal, low to high or from normal to high], categorized no change [value stays in the same reference range], categorized decrease [shift from high to normal, high to low or from normal to low]).

The following list of parameters will be summarized using descriptive statistics and for the shift table.

 Table 21
 Laboratory Parameters for Descriptive Statistics and Shift Table

| Lab Panel | <b>Analysis Time Point</b> | Parameter |
|---|---|---|
| Hematology and | Baseline | Hemoglobin |
| Coagulation | | Hematocrit |
| | <u>Treatment period</u> | Erythrocytes (Red blood cell [RBC]) |
| | Week 2, | Leukocytes (White blood cell [WBC]) |
| | Week 4, | Differential WBC |
| | Week 8, | Platelets |
| | | PT and INR |
| | Follow-up | MCV |
| | Week 10 | MCH |
| | | Reticulocytes |
| Biochemistry | Baseline | Sodium |
| | | Potassium |
| | <u>Treatment period</u> | Calcium |
| | Week 2, | Chloride |
| | Week 4, | Magnesium |
| | Week 8, | Glucose |
| | | Creatine Kinase |
| | Follow-up | Creatinine |
| | Week 10 | Alkaline Phosphatase (ALP) |
| | | Lactate dehydrogenase (LDH) |
| | | Aspartate transaminase (AST) |
| | | Alanine transaminase (ALT) |
| | | Gamma glutamyl transpeptidase (GTT) |
| | | Total bilirubin (direct and indirect) |
| | | Total protein |
| | | Albumin |
| | | Total cholesterol |
| | | Triglycerides |
| | | Uric Acid |
| | | Blood Urea Nitrogen (BUN) |
| | | Inorganic phosphate |

All laboratory measurements, including the derived outcomes (change from baseline and flagging of abnormal value with high and low) will be presented in the listing. Urinalysis will be listed only.

## 7.5.3.1 Liver Enzymes and Total Bilirubin

The following potentially clinically significant (PCS) criteria for liver tests – defined as Alkaline Phosphatase (ALP), Alanine Transaminase (ALT), total bilirubin (TBL), Aspartate Transaminase (AST), International Normalized Ratio (INR) and their combination are defined.

Table 22 Potentially Clinically Significant Criteria for Liver Enzymes and Total Bilirubin

| Parameter | Criteria |
|---|---|
| ALT | > 3xULN |
| | > 5xULN |
| | > 10xULN |
| | > 20xULN |
| AST | > 3xULN |
| | >5xULN |
| | > 10xULN |
| | > 20xULN |
| ALT or AST | > 3xULN |
| TBL | >2xULN |
| INR | > 1.5 (Ratio) |
| ALP | > 1.5xULN |
| ALT and/or AST AND TBL (*) | (ALT and/or AST > 3xULN) and TBL > 2xULN |
| ALT and/or AST AND | (ALT and/or AST > 3xULN) and (TBL > 2xULN and/or INR > 1.5 |
| TBL and/or INR <sup>(*)</sup> | |

<sup>(\*)</sup> Combination of values measured from the samples collected on the same day.

The number and percentage of subjects with PCS values in liver enzyme and total bilirubin tests using the subject's highest value during the double-blind treatment period will be presented by treatment group. Another summary will be created using the subject's highest value during the follow-up period.

In addition to the above summaries the following data will be presented graphically by treatment group:

- Scatter plot of maximum values for ALT or AST and TBL during the double-blind treatment period and follow-up period with ALT or AST values on x-axis and TBL values on y-axis [Senior, 2014], and
- Individual display of liver enzymes and TBL for selected subjects experiencing potentially clinically significant criteria of ALT > 3xULN or AST > 3xULN or TBL > 2xULN during double-blind treatment period or follow-up period.

## 7.5.3.2 Potentially Clinically Significant Laboratory Criteria

Potentially clinically significant laboratory criteria for other laboratory variables are provided in Section 10.3 Appendix 3: Potentially Clinically Significant Laboratory Criteria The number and percentage of subjects with PCS values using the subject's highest and/or lowest value (depending on the direction of interest) during the double-blind treatment period will be presented by treatment group. Another summary will be created using the subject's highest and/or lowest value (depending on the direction of interest) during the follow-up period.

## 7.5.4 Vital Signs

The baseline visit is the last measurement taken prior to the first dose of study drug.

Supine (average)/resting vital signs (SBP, DPB and pulse rate) will be summarized using mean, SD, minimum, maximum and median by treatment group and visit (Baseline, Day 1 2-hours post-dose, Week 2, Week 4, Week 8/EOT, Week 10). Additionally, a within-subject change will be calculated per visit as the post-baseline measurement minus the baseline measurement and summarized by treatment group and visit. Section 7.11.5.3 describes the derivation of visit windows for vital signs.

Standing vital signs (SBP, DPB and pulse rate) will be summarized using mean, SD, minimum, maximum and median by treatment group and visit (Baseline, Day 1 2-hours post-dose, Week 8 / EOT). Additionally, a within-subject change will be calculated per visit as the post-baseline measurement minus the baseline measurement and summarized by treatment group and visit.

Table 23 describes PCS criteria for vital signs. The number and percentage of subjects with PCS values in vital signs using the subject's worst value during double-blind treatment period will be presented by each treatment group. The summary will include all vital signs at both scheduled and unscheduled visits. It will include resting and orthostatic (supine [average] and standing) vital signs. For criteria comparing with baseline, vital signs at standing will be compared with vital signs at standing and vital signs at supine (average)/resting will be compared with vital signs at supine (average)/resting.

Another summary will be created using the subject's worst value (resting vital signs only) during the follow-up period.

| Table 22 | Datantialler | Climinaller | Ciarrificant | Cuitania | for Vital Ciana |
|---|---|---|---|---|---|
| Table 23 | Potentiany | Cillicaliv | Significant | Criteria i | for Vital Signs |

| Vital Sign Parameter | Criteria | Worst Value |
|---|---|---|
| SBP | • <90 mmHg | Lowest |
| | • Decrease of $\geq$ 20 mmHg from baseline | Lowest |
| | • >180 mmHg | Highest |
| | • Increase of ≥20 mmHg from baseline | Highest |
| DBP | • <40 mmHg | Lowest |
| | • Decrease of $\geq$ 20 mmHg from baseline | Lowest |
| | • >100 mmHg | Highest |
| | • Increase of ≥ 20 mmHg from baseline | Highest |
| Pulse rate | • <50 bpm | Lowest |
| | • Decrease of $\geq$ 20 bpm from baseline | Lowest |
| | • <50 bpm and decrease of ≥ 20 bpm from baseline (*) | Lowest |
| | • >100 bpm | Highest |
| | • Increase of $\geq 20$ bpm from baseline | Highest |
| | • >100 bpm and increase of $\geq$ 20 bpm from baseline (*) | Highest |

<sup>(\*)</sup> Combination of values from the same time point.

Table 24 describes orthostatic outlier criteria for vital signs. The number and percentage of patients with orthostatic outlier values in vital signs will be presented by each treatment group at each post-baseline time point. For the overall during the double-blind treatment period, a subject's largest drop during that period will be used. The summary will also include results for the number and percentage of subjects where orthostatic challenge test lead to clinically significant results or symptoms.

**Sponsor:** Astellas Pharma Global Development, Inc. (APGD)

ISN/Protocol 8062-CL-0101

| Table 27 Orthostalic Outlier Criteria for Vitar Sign | Table 24 | Orthostatic Outlier Criteria | for V | Vital Sign |
|---|---|---|---|---|
|---|---|---|---|---|

| <b>Analysis Time Point</b> | Vital Sign Parameter | Criteria |
|---|---|---|
| Treatment period | Orthostatic SBP | ≥ 20 mmHg decrease from average supine value |
| | Orthostatic DBP | ≥10 mmHg decrease from average supine value |
| Day 1 2-hours post-dose, | Orthostatic Challenge | ≥20 mmHg decrease from average supine value for |
| Week 8 / EOT, | Test | orthostatic SBP |
| Double-blind treatment | | OR |
| period | | ≥10 mmHg decrease from average supine value for |
| | | orthostatic DBP |
| | Orthostatic Pulse rate | ≥20 bpm increase from average supine value |

## 7.5.5 Electrocardiograms

The baseline visit is the last measurement taken prior to the first dose of study drug.

The number and percentage of subjects with normal, not clinically significant abnormal, and clinically significant abnormal results as assessed by investigator for the 12-lead ECG will be tabulated by treatment group at each treatment visit and time point (Baseline, Week 8, EOT and Week 10).

Number and percent of subjects with 12-lead ECG abnormalities as well as number and percent of subjects whose 12-lead ECG reading changed from normal at baseline to abnormal will be tabulated by treatment group at each treatment visit and time point (Baseline, Week 8, EOT and Week 10)

A shift table of the finding at baseline ('normal', 'abnormal - not clinically significant' and 'abnormal - clinically significant') to the worst finding during the double-blind treatment period and follow-up period will be presented by treatment group.

#### 7.5.6 Physical Examination Findings

Physical examination findings will be listed by treatment group.

## 7.5.7 Columbia Suicide Severity Rating Scale

Number and percentage of subjects in each of the categories of C-SSRS described in Section 6.2.5 will be summarized at each analysis time point (Baseline, Week 2, Week 4, Week 8, EOT and Week 10) by treatment group. For each analysis time point, if a subject answers "yes" to more than one question within a category, the worst finding will be used.

For the overall during the double-blind treatment period and the overall during the follow-up period, a subject's worst finding during that period will be used.

All C-SSRS assessments will be listed only for subjects with at least one event of suicidality (suicidal ideation and/or suicidal behavior).

## 7.5.8 Pregnancies

A detailed listing of all pregnancies will be provided.

# 7.6 Analysis of Pharmacokinetics

PK assessments will only be performed in subjects treated with ASP8062. Summary tables of PK concentration will be provided for Day 1 (1-4 hours post-dose) and by sampling
timepoint (pre-dose, 1-4 hours post dose and >4 hours post dose) across Weeks 2, 4 and 8/EOT combined (see table below). Descriptive statistics will include n [number of samples], mean, standard deviation, minimum, median, maximum, coefficient of variation and geometric mean.

PK Summary Table Schema

| Week 1 | Weeks 2, 4, 8/EOT | | |
|---|---|---|---|
| 1-4 hours post dose | Pre-dose | 1-4 hours post dose | >4 hours post dose |

A listing of sample times and concentrations will be provided.

#### 7.7 Analysis of Pharmacodynamics

Not applicable.

## 7.8 Subgroups of Interest





## 7.9 Other Analyses

No additional analyses are planned.

#### 7.10 Interim Analysis (and Early Discontinuation of the Clinical Study)

Two interim analyses for futility based on the primary efficacy endpoint will be conducted. The timing of these analyses will be at approximately 35% and 55% of all subjects with Week 8/EOT data. The plan for the interim analysis may be modified based on speed of recruitment. These analyses will be conducted by an Astellas statistician, with results reviewed by an Astellas IDMC. The Astellas statistician and other members of the Astellas IDMC are external to the study team. No one within the study team will be unblinded to the treatment allocation or interim results. Details of the interim analysis procedure, steps to maintain treatment blind in the study team and criteria for stopping the study will be described in an IAP.

# 7.11 Handling of Missing Data, Outliers, Visit Windows, and Other Information

#### 7.11.1 Missing Data

As a general principle, no imputation of missing data for other variables will be done. Exceptions are the onset date of AE, start and stop dates of non-medication therapy, start and stop dates of previous and concomitant medication, onset date of FM symptoms, date of FM diagnosis and first/last dose date of double-blind study drug. In the listings of AEs, non-medication therapy, previous and concomitant medication and onset date of FM symptoms, diagnosis of FM, the first dose/last dose date of double-blind study drug will present the actual partial dates; imputed dates will not be shown.

For one of the sensitivity analyses for the primary efficacy endpoint and one of the sensitivity analysis for the FIQR secondary endpoint, multiple imputation will be used to impute missing data, using a discontinuation reason-based approach as described in Section 7.4.1.2 For analyses of selected efficacy endpoints, mBOCF, BOCF and/or LOCF will be used to impute the missing data. More details are described in Section 6.1 and Section 7.4

#### **Imputation of Adverse Event Onset Date**

For AEs, a missing or incomplete onset date will be imputed according to the following conventions:

If an onset date is missing or only the year is known, the imputed onset date will be the <u>latest</u> of the following non-missing dates:

- First dose date of double-blind study drug
- Randomization date + 1 day

If only the month and year is known for onset date, set the surrogate onset date to the first day of that month and then apply the following rules:

1. If the month and year of the onset date is prior to the month and year of the first dose of double-blind study drug, then the surrogate onset date will be the imputed onset date.

2. If the month and year of the onset date is on or after the month and year of the first dose of double-blind study drug, then the imputed onset date will be the <u>latest</u> of the following non-missing dates:

- First dose date of double-blind study drug
- Randomization date + 1 day
- Surrogate onset date

If the imputed onset date is after a complete adverse event end date, the imputed onset date will be the same as the complete adverse event end date.

#### **Imputation of Adverse Event End Date**

If only the day is missing for end date, set the surrogate end date to the last day of the month.

If the day and the month are missing for end date, set the surrogate end date month to December and set the day to the last day of the month (31).

If the year or the entire end date is missing, end date will not be imputed.

If an AE end date has been imputed, then apply the following rule:

1. If this imputed date falls after the end of participation in the study, then the surrogate end date will be set to the date of end of participation.

If the AE is ongoing (outcome is "NOT RECOVERED/NOT RESOLVED" or "RECOVERING/RESOLVING") then the end date will remain missing.

# <u>Imputation of Start and Stop Dates of Non-Medication Therapy and Previous and Concomitant Medication Dates</u>

For Non-Medication Therapy and Previous and Concomitant Medications, a missing or incomplete start and stop dates will be imputed according to the following conventions:

If start date is missing or partial:

- if month is missing, use January
- if day is missing, use the first day of the month under consideration
- if year is missing, use year of the informed consent date
- if entire date is missing, use informed consent date

If stop date is missing or partial and medication or therapy is not ongoing:

- if month is missing, use December
- if day is missing, use the last day of the month under consideration
- if year or the entire date is missing, set to December 31<sup>st</sup>, 2099

If the imputed start date is after the stop date, then the imputed start date will be one day prior to the stop date.

If the medication or therapy is ongoing, the stop date will remain missing.

#### Missing Onset Date of FM Symptoms and Date of FM Diagnosis

An incomplete onset date of FM Symptoms or date of FM diagnosis will be imputed according to the following conventions:

• Missing day, but month and year are present: the day will be imputed as the 15<sup>th</sup> day of the month.

SAP Final Version 2.0

- Missing day and month, but year is present: the day and month will be imputed as 30 June of the year.
- Missing year, but day and month are present: No imputations will occur, and the subject will be excluded from all summaries related to time since FM symptoms and diagnosis.
- Missing day, month and year: No imputations will occur, and the subject will be excluded from all summaries related to time since FM symptoms and diagnosis.
- If any such imputed date falls after the informed consent date, then the onset date will be taken as equal to the informed consent date.

#### **Imputation of Study Drug Start Date Double-Blind Treatment Period**

For subjects who are randomized to double-blind study drug, the first dose date of double-blind study drug will be imputed if both of the following criteria are met:

- There is a missing or partial date for the first dose of double-blind study drug AND
- The number of tablets dispensed does not equal the number of tablets returned (including missing values).

If the first dose date of double-blind study drug is missing or partial, the first dose date of double-blind study drug is defined as the non-missing dispense date at randomization.

#### **Imputation of Study Drug End Date Double-Blind Treatment Period**

For subjects who are randomized to double-blind study drug, the last dose date of double-blind study drug will be imputed if both of the following criteria are met:

- There is a missing or partial date for the last dose of double-blind study drug AND
- The number of tablets dispensed does not equal the number of tablets returned (including missing values).

If only the day is missing for the last dose date of double-blind study drug, the last day of the month under consideration will be used.

If the month and/or year are missing for the last dose date of double-blind study drug, then the <u>latest</u> of the following non-missing dates will be used:

- 11. last dispense date + 1 day OR
- 12. the date of the last vital sign measurement during the double-blind treatment period OR
- 13. 3.the date of the first dose of double-blind study drug in the double-blind treatment period + 1 day

SAP Final Version 2.0

ISN/Protocol 8062-CL-0101

#### **7.11.2 Outliers**

All values will be included in the analyses.

#### 7.11.3 Values Below Limit of Quantification (BLOQ)

For quantitative laboratory variables, values recorded as "<X" or "<=X" or ">Y" or ">=Y" will be imputed by "X" and "Y" respectively for descriptive statistics. This will be documented in a footnote to all summary tables and all output where such a replacement was performed.

ASP8062 plasma concentrations that are below the limit of quantification (BLOQ) will be set to 0 for calculating descriptive statistics.

#### 7.11.4 Visit Windows for Efficacy Variables

#### 7.11.4.1 Duplicate Values

For daily average pain scores assessed by NRS any data captured in the e-diary up to 2am in the morning of the following day will be assigned to the previous day in the derivation of Study Day (Section 7.1).

For all efficacy variables (either recorded in the e-diary or the tablet device), if more than one value is measured/recorded on the same Study Day, then the first of the values will be used. This should be applied before implementing the visit windows as described in Section 7.11.4.3

#### 7.11.4.2 Post Dosing Efficacy Observations

For efficacy variables, observations will not contribute to the efficacy analyses during the treatment period if the subject's last dose of double-blind study drug is as follows:

Any diary days or non-diary days which are > 4 days after the last dose of double-blind study drug will not be included in the analysis related to on-treatment time points and the EOT time point. This should be applied before implementing the visit windows in Section 7.11.4.3

#### 7.11.4.3 Visit Windows

Subjects do not always adhere strictly to the visit timing in the protocol. Therefore, the designation of time points will be based on Study Day and Follow-Up Day (as defined in Section 7.1) rather than the nominal visit recorded in the eCRF.

To assign a measurement to a Week t during the double-blind treatment period, the first step consists of selecting all measurements falling within the double-blind treatment period as defined above. To further determine the Week t measurement, mutually exclusive relative day windows are used.

These day windows are defined to provide derived time points that correspond to the post baseline time points specified in the protocol.

Table 26 provides day windows for daily average pain scores assessed by NRS and rescue medication data.

Table 26 provides day windows for daily average pain scores assessed by NRS and rescue medication data.



Table 27 Day Windows: FMSD Questionnaire

| Analysis Time Point | Visit Window (Day) |
|---|---|
| Baseline | Study days -6 to 1 |
| Week 1 | Study days 3 to 8 |
| Week 2 | Study days 9 to 15 |
| Week 3 | Study days 16 to 22 |
| Week 4 | Study days 23 to 29 |
| Week 5 | Study days 30 to 36 |
| Week 6 | Study days 37 to 43 |
| Week 7 | Study days 44 to 50 |
| Week 8 | Study days 51 to 57 |
| EOT | Study day 3 to 57, where post-baseline data from the last 7 calendar days on |
| | or prior to the last FMSD scores will be used. If there is no post baseline |
| | data available EOT will be imputed using the baseline measurement. |
| Week 10 | Follow up days 8 to 14 |



| Table 29 Day V | Vindows: HADS, | |
|----------------------|------------------|------------------------|
| Analysis Time point | Target Day | Visit Window (Day) |
| Week 8 | Study day 57 | Study day 44 to 71 |
| Week 10 <sup>b</sup> | Follow-up day 14 | Follow-up days 5 to 28 |

Baseline is defined as the last assessment on or prior to the first dose day (Day 1) of double-blind study drug.

For efficacy variables recorded in the e-diary (NRS questionnaire, rescue medication and , the following rule will apply:



For efficacy variables recorded in the tablet device, the following rule will apply:

• If a subject has more than one time point with a measurement included within a window, the assessment closest to the target day will be used. In case of ties between observations located on different sides of the scheduled day, the later assessment will be used. In case of ties located on the same side of the scheduled day (i.e. more than one value for the same day), the first value will be used.

#### 7.11.5 Visit Windows for Safety Variables

#### 7.11.5.1 Duplicate Values

For safety laboratory data and vital signs (apart from orthostatic vital signs)- if more than one value is reported on the same day, then the mean of the values will be used. This needs to be done before creating the analysis time points.

For orthostatic vital signs the average of the triplicates for supine measurements must be calculated first. If there are more than one set of triplicate measurements at a timepoint, both orthostatic values will be calculated and used in the PCS vital sign and orthostatic outlier table. If there are more than one orthostatic measurements in the same time window, the later one will be used for the change from baseline calculation.

#### 7.11.5.2 Post Dosing Safety Observations

For safety variables, observations will not contribute to the safety analyses during the treatment period if the subject's last dose of double-blind study drug is as follows:

Any days which are > 4 days after the last dose of double-blind study drug will not be included in the analysis related to on-treatment time points and the EOT time point. This needs to be done before creating the analysis time points.

#### 7.11.5.3 Visit Windows

Table 30 provides day windows for safety laboratory variables, vital sign variables and C-SSRS. Table 31 provides day windows for the categorical ECG assessment.

Table 30 Day Windows: Laboratory, Vital Sign Variables and C-SSRS

| <b>Analysis Time Point</b> | Target Day | Visit Window (Day) |
|---|---|---|
| Week 2 | Study day 15 | Study days 2 to 22 |
| Week 4 | Study day 29 | Study days 23 to 43 |
| Week 8 | Study day 57 | Study days 44 to 71 |
| EOT <sup>a</sup> | Not applicable | Study day 2 to Follow-up day 4 |
| Double-blind treatment period <sup>b</sup> | Not applicable | Study day 2 to Follow-up day 4 |
| Week 10 <sup>c</sup> | Follow up day 14 | Follow-up days 5 to 28 |
| Follow-up period <sup>d</sup> | Not applicable | Follow-up day 5 onwards |

Baseline is defined as the last assessment on or prior to the first dose day (Day 1) of double-blind study drug.

Table 31 Day Windows: Categorical ECG Assessment

| <b>Analysis Time Point</b> | Target Day | Visit Window (Day) |
|---|---|---|
| Week 8 | Study day 57 | Study days 44 to 71 |
| EOT <sup>a</sup> | Not applicable | Study day 2 to Follow-up day 4 |
| Double-blind treatment period <sup>b</sup> | Not applicable | Study day 2 to Follow-up day 4 |
| Week 10 | Follow-up day 14 | Follow-up days 5 to 28 |
| Follow-up period | Not applicable | Follow-up day 5 onwards |

Baseline is defined as the last assessment on or prior to the first dose day (Day 1) of double-blind study drug.

For safety variables, the following rules will apply:

- 1. For laboratory and vital sign variables, if a subject has more than one visit with a measurement included within a window, the assessment closest to the target day will be used. In case of ties between observations located on different sides of the scheduled day, the later assessment will be used. In case of ties located on the same side of the target day (i.e., more than one value for the same day), the mean of the values will be used.
- 2. For the categorical ECG assessment, if a subject has more than one result with a measurement included within a window, the assessment closest to the target day will be used. In case of ties between observations located on different sides of the target day, the later assessment will be used in the analyses. In case of ties located on the same side

<sup>&</sup>lt;sup>a</sup> EOT value is the last available non-missing post-baseline measurement within the visit window. Vital signs will also include Day 1 2 hours post-dose.

<sup>&</sup>lt;sup>b</sup>Only applicable to potentially clinically significant laboratory parameters, potentially clinically significant vital signs, orthostatic outlier vital signs and C-SSRS. Vital signs will also include Day 1 2 hours post-dose.

<sup>&</sup>lt;sup>c</sup>Orthostatic vital signs are not captured at Week 10.

<sup>&</sup>lt;sup>d</sup>Only applicable to potentially clinically significant laboratory parameters, potentially clinically significant vital signs and C-SSRS.

<sup>&</sup>lt;sup>a</sup> EOT value is the last available non-missing post-baseline measurement within the visit window.

- of the scheduled day (i.e., more than one value for the same day), the worst-case parameter value (where 'abnormal clinically significant' is considered worse than 'abnormal not clinically significant', which in turn are both considered worse than 'normal').
- 3. For the C-SSRS, if a subject answers 'yes' to more than one question within a window, the worst-case response (within a category) will be used irrespective of whether this is closest to the target day.

#### 7.11.6 Pooling Sites Algorithm

Approximately 178 subjects will be enrolled in approximately 35 sites. When "center" is included as a factor in a statistical model, sites that have less than 10 FAS subjects in total will be identified and then combined for statistical analysis purpose according to the following algorithm:

- Step 1. Divide the sites into 2 groups with Group 1 including all sites that have at least 10 FAS subjects in total and Group 2 including all remaining sites. Sort each group in ascending order by total sample size and site number.
- Step 2. Starting at the top of the Group 2 list (i.e., the first site with the smallest total sample size), combine the minimum number of sites required to achieve a "study site" that has at least 10 FAS subjects in total. Continue forming "center" in this manner until all Group 2 sites have been grouped or it is no longer possible to form a "center" with at least 10 FAS subjects in total.
- Step 3. If there is a site (or several sites) left after step 2, combined the site(s) with the last pooled site that is created. For the situation where no previous pooled site is created, combine the site(s) with the first site on the sorted Group 1 list.

Pooled sites will be assigned names PoolSite01, PoolSite02, etc.

For all sites that have been combined into pooled sites, the assigned pooled site will be used instead of the original site identification in all statistical models that include "center" as a factor. However, the original site identification will be used in all summaries of subject disposition or discontinuation by site and in all data listings.

#### 8 DOCUMENT REVISION HISTORY

| <u>Version</u> | <u>Date</u> | Changes | Comment/rationale for change |
|---|---|---|---|
| 1.00 | 05-APR-2017 | NA | Document finalized |
| 2.0 | 19-Apr-2018 | Section 5.2.1 Table 2:<br>Updated criteria to | Typographical errors. |
| | | criterion where appropriate. | Additional text included for clarification to match classification specification |
| | | Additional text included for FIQR inclusion criteria: 'Inclusion | |
| | | criterion #12 is No<br>and/or FIOR pain item | |

| Version | <u>Date</u> | Changes | Comment/rationale for change |
|---|---|---|---|
| | | score < 4 at Screening.' | |
| 2.0 | 19-Apr-2018 | Section 6.1: Additional sentence added: 'For FIOR. PGIS, and HADS baseline is defined as the last assessment on or prior to the first dose day (Day 1) of double-blind study drug. | Clarification of derivation of baseline for questionnaires captured on the tablet at site. |
| 2.0 | 19-Apr-2018 | | |
| 2.0 | 19-Apr-2018 | | |
| 2.0 | 19-Apr-2018 | | |

| Version | <u>Date</u> | Changes | Comment/rationale for change |
|---|---|---|---|
| 2.0 | 19-Apr-2018 | Section 6.1.3 Table 9: | Additional text included to define the |
| | 1 | Total Number of days | denominator for each week (Total number of |
| | | replaced with | days) for subjects who discontinue early or |
| | | 'Minimum of (upper | who come in early for their last visit (but |
| | | bound of the time | within the designated window in the |
| | | window, last assessment | protocol.) |
| | | day from e-dairy data) – | |
| | | lower bound of the time window + 1' | |
| 2.0 | 19-Apr-2018 | Section 6.4.7: | Extra clarification regarding derivation of |
| 2.0 | 19-Api-2016 | Additional sentences | CMSI total score and definition of baseline. |
| | | added to the end of this | Civisi total score and definition of baseline. |
| | | section: | |
| | | 'The CMSI total score at | |
| | | baseline will be | |
| | | calculated and ranges | |
| | | from 0 to 39 for males | |
| | | and 0 to 41 for females. | |
| | | Baseline is defined as | |
| | | the last assessment on or | |
| | | prior to the first dose<br>day (Day 1) of double- | |
| | | blind study drug.' | |
| 2.0 | 19-Apr-2018 | Section 7.1: | Extra clarification regarding the number of |
| 2.0 | 1) 11pt 2010 | Additional sentences | subjects which will be presented in summary |
| | | added to the end of the | tables. |
| | | following paragraph: | |
| | | 'Summaries based on | |
| | | FAS and PPS (e.g. | Significance level added for 2-sided p-values. |
| | | disposition, baseline and | |
| | | efficacy data) will be | |
| | | presented by planned treatment group, unless | |
| | | specifically stated | |
| | | otherwise. Safety | |
| | | analysis and other | |
| | | summaries based on | |
| | | SAF will be presented | |
| | | by actual treatment | |
| | | received. For | |
| | | summaries which | |
| | | present both absolute values over time and | |
| | | change from baseline | |
| 1 | | values over time the | |
| | | number of subjects | |
| 1 | | used to calculate the | |
| | | descriptive statistics | |
| 1 | | will be those who have | |
| 1 | | non-missing data at | |
| | | each analysis visit and | |
| | | at baseline. For | |
| | | endpoints which include mBOCF, | |
| | | LOCF or mLOCF | |
| | | LOCT OF INLOCE | |

| <u>Version</u> | <u>Date</u> | <u>Changes</u> | Comment/rationale for change |
|---|---|---|---|
| | | imputation the descriptive statistics will be calculated after the imputation has been performed. | |
| | | Unless otherwise specified, statistical comparisons will be made using one-sided tests at the α=0.05 significance level and two-sided 90% confidence intervals (CIs) will be presented when applicable. When two-sided p-values are presented statistical comparisons will be made using an α=0.1 | |
| 2.0 | 19-Apr-2018 | significance level. Section 7.2.4: Additional paragraph added: All previous medications for taken for any pain prior to the baseline diary run-in; all previous medications taken for any pain during baseline diary run-in; all concomitant medications taken for any pain during the double blind treatment period and all concomitant medications taken for any pain during the follow-up period will also be summarized by preferred WHO name by treatment group and 'Total' over all treatment groups. | Description of extra summaries of previous medications and concomitant medications for any pain added. |

| Version | <u>Date</u> | Changes | Comment/rationale for change |
|---|---|---|---|
| 2.0 | 19-Apr-2018 | Section 7.2.3.3, Table 14: Additional group added to each of CMSI total score and Footnote regarding definition of cut-points for CMSI total score and updated. | Decision made to split CMSI total score into three groups: |
| 2.0 | 19-Apr-2018 | Section 7.4.1.1: In the description of the MMRM model the text 'baseline mean daily average pain score-bytreatment interaction' has been replaced by 'baseline mean daily average score-by-time interaction' and subject as a random effect has been removed from the model | Typographical error 'treatment' replaced with 'time'. Subject as a random effect has been removed from model due to issues with convergence. |
| 2.0 | 19-Apr-2018 | | |
| 2.0 | 19-Apr-2018 | | |

| Version | <u>Date</u> | Changes | Comment/rationale for change |
|---|---|---|---|
| 2.0 | 19-Apr-2018 | | |
| 2.0 | 19-Apr-2018 | | |
| 2.0 | 19-Apr-2018 | | |
| 2.0 | 19-Apr-2018 | Section 7.5.1.3: Text updated so that AEs with missing severity will be imputed with worst severity, i.e severe rather than treated as missing. | Updated to comply with latest version of Astellas standards |

| Version | Date | Changes | Comment/rationale for change |
|---|---|---|---|
| 2.0 | 19-Apr-2018 | Section 7.5.3: Bullet point describing summary shifts of laboratory parameters so that 'low to high' is included as a categorized increase and 'high to low' is included as a categorized | Study team feedback provided that these extra conditions should be included in these definitions. |
| 2.0 | 19-Apr-2018 | decrease. Section 7.8.1: Text updated to describe updates to the cut-points being used to split the CMSI total score, into subgroups. | Decision made to split CMSI total score into three groups; |
| 2.0 | 19-Apr-2018 | Section 7.11.4.3: Tables 21 and 22 Imputation of EOT updated to specify that baseline is carried forward when there are no measurements post baseline. | Extra clarification regarding imputation at EOT timepoint provided for NRS, FIQR, PGIS, PGIC HADS, and Definition of baseline provided for PGIS, and |
| | | Tables 23 and 24 Extra footnote providing the definition of baseline and imputation of EOT when there are no post-baseline measurements added. | |
| 2.0 | 19-Apr-2018 | Section 7.11.5.3:<br>Extra footnote providing<br>definition of baseline<br>added to Tables 25 and<br>26. | Extra clarification regarding definition of baseline for laboratory parameters, vital signs variables, C-SSRS questionnaire and ECG assessments. |
| 2.0 | 19-Apr-2018 | Section 7.11.5.3, Table 30. Footnote clarifying that vital signs are also collected on study day 1 at 2 hours post-dose | Updated to specify that vital signs are also collected on study day 1 at 2 hours post-dose |
| 2.0 | 19-Apr-2018 | Appendix 10.1: MedDRA version updated to 20.0. List of Lower Level Terms updated to reflect update to MedDRA v2.0. Lower Level Codes added to table. | Table updated to reflect change to MedDRA v20.0 |
| 2.0 | 19-Apr-2018 | Appendix 10.2:<br>MedDRA version | Table updated to reflect change to MedDRA v20.0 |

| Version | <u>Date</u> | Changes | Comment/rationale for change |
|---|---|---|---|
| | | updated to 20.0. List of<br>Lower Level Terms<br>updated to reflect update<br>to MedDRA v2.0.<br>Lower Level Codes<br>added to table. | |
| 2.0 | 19-Apr-2018 | Section 6.1, 7.2 and 7.4: "FIQR physical function" was changed to "FIQR function" wherever it was mentioned. | Typographical error. |

#### 9 REFERENCES

- Carpenter JR, Roger JH & Kenward MG. Analysis of longitudinal trials with protocol deviation: a framework for relevant, accessible, assumptions, and inference via multiple imputation. Journal of Biopharmaceutical Statistics. 2013;23(6):1352-1371.
- ICH Harmonized Tripartite Guideline E 3. Structure and Content of Clinical Study Reports, November 1995. (www.ich.org; Guidelines; "Efficacy" Topics).
- ICH Harmonized Tripartite Guideline E 9. Statistical Principles for Clinical Trials, February 1998. (www.ich.org; Guidelines; "Efficacy" Topics).
- O'Kelly M & Ratitch B. Clinical Trials with Missing Data: A Guide for Practitioners. Statistics in Practice (2014):189 190.
- Senior JR. Evolution of the Food and Drug Administration Approach to Liver Safety Assessment for New Drugs: Current Status and Challenges. Drug Safety (2014) 37 (Suppl 1): S9–S17.

### 10 APPENDICES

## **10.1** Appendix 1: Drug Abuse Related Adverse Events

Abuse related adverse events of interest (MedDRA 20.0) that are explicitly referenced in the 2010 draft guidance

| System | Higher Level | Higher | Preferred | <b>Lowest Level Term</b> | Lower Level Code |
|---|---|---|---|---|---|
| Organ Class | GT | Level Term | term | | |
| Psychiatric | Mood | Emotional | Euphoric | Euphoria | 10015533 |
| disorders | | and mood | Mood | Euphoric | 10015534 |
| | disturbances | disturbances | | Euphoric mood | 10015535 |
| | NEC | NEC | | Exaggerated well- | 10015584 |
| | | | | being | |
| | | | | Feeling high | 10016333 |
| | | | | Felt high | 10016382 |
| | | | | High | 10020044 |
| | | | | High feeling | 10020063 |
| | | | | Hyperthimic | 10020847 |
| | | | | Hyperthimic state | 10020849 |
| | | | | Laughter | 10024042 |
| | | | | Mood elevated | 10027949 |
| | | | Mood altered | Affect alteration | 10054199 |
| | | | | Affect altered | 10001439 |
| | | | | Altered mood | 10001850 |
| | | | | Bad mood | 10004064 |
| | | | | Mood alteration | 10027937 |
| | | | | NOS | |
| | | | Mood altered | 10027940 | |
| | | | | Mood change | 10027941 |
| | | Affect | Inappropriate | Elation | 10014339 |
| | | alterations | affect | inappropriate | |
| | | | | Exhilaration | 10015672 |
| | | | | inappropriate | |
| | | | | Exhilaration | 10015673 |
| | | | Feeling hap | inappropriate | |
| | | | | Feeling happy | 10016332 |
| | | | | inappropriately | |
| | | | | Inappropriate affect | 10021588 |
| | | | | Inappropriate crying | 10021589 |
| | | | | Inappropriate elation | 10021592 |
| | | | | Inappropriate | 10021593 |
| | | | | exhilaration | |
| | | | | Inappropriate | 10021595 |
| | | | | laughter | |
| | | | | Inappropriate mood | 10021596 |
| | | | | elevation | |
| | | | | Mood elevation | 10027950 |
| | | | | inappropriate | |

| System<br>Organ Class | Higher Level<br>GT | Higher<br>Level Term | Preferred<br>term | Lowest Level Term | Lower Level Code |
|---|---|---|---|---|---|
| Psychiatric | Disturbances | Perception | Hallucination | Drug-induced | 10013761 |
| disorders | in thinking | disturbances | | hallucinosis | |
| | and | | | Hallucinating | 10019062 |
| | perception | | | Hallucination | 10019063 |
| | 1 1 | | | Hallucination NOS | 10019066 |
| | | | | Hallucinations | 10019077 |
| | | | | Hallucinations | 10019078 |
| | | | | aggravated | 10017070 |
| | | | | Kinesthetic | 10023450 |
| | | | | hallucination | 10025450 |
| | | | | Organic hallucinosis | 10031079 |
| | | | | syndrome | 10031077 |
| | | | | Pseudohallucination | 10066297 |
| | | | | Sensory | 10040028 |
| | | | | hallucinations | 10040026 |
| | | | | Stump hallucination | 10042263 |
| | | | Hallucination, | Auditory | 10042203 |
| | | | auditory | hallucinations | 10003783 |
| | | | auditory | Hallucination | 10019064 |
| | | | | auditory | 10019004 |
| | | | | Hallucination, | 10019070 |
| | | | | | 10019070 |
| | | | | auditory<br>Verbal | 10069415 |
| | | | | hallucinations | 10009413 |
| | | | Hallucination, | Hallucination visual | 10019068 |
| | | | visual | Hallucination with | 10019008 |
| | | | visuai | color | 10033327 |
| | | | | Hallucination with | 10019069 |
| | | | | | 10019069 |
| | | | | colour | 10019075 |
| | | | | Hallucination, visual | 10019073 |
| | | | | 77' 1 | 10047570 |
| | | | | Visual | 10047570 |
| C 1 | C 1 | F. din | P I'm | hallucinations | 10012767 |
| General | General | Feelings and | Feeling drunk | Drunk-like effect | 10013767 |
| disorders and administratio | system | sensations<br>NEC | | Drunkenness feeling | 10013769 |
| n site | NEC NEC | NEC | | Of<br>Facility of decorate | 1001(220 |
| conditions | NEC | | P. die. | Feeling drunk | 10016330 |
| Conditions | | | Feeling abnormal | Cotton wool in head | 10011221 |
| | | | abnormai | Feeling abnormal | 10016322 |
| | | | | Feeling bad | 10016324 |
| | | | | Feeling dazed | 10050462 |
| | | | | Feeling floating | 10016331 |
| | | | | Feeling lifeless | 10016340 |
| | | | | Feeling miserable | 10016342 |
| | | | | Feeling stoned | 10070679 |
| | | | | Feeling strange | 10016366 |
| | | | | Feeling weightless | 10016372 |
| | | | | Feels awful | 10016375 |
| | | | | Feels bad | 10016376 |
| | | | | Feels poorly | 10016377 |
| | | | | Felt like a zombie | 10016384 |
| | | | | Floating feeling | 10016782 |

| System | Higher Level | Higher | Preferred | <b>Lowest Level Term</b> | Lower Level Code |
|---|---|---|---|---|---|
| Organ Class | GT | Level Term | term | | |
| | | | | Foggy feeling head | 10016876 |
| | | | | Funny episode | 10017552 |
| | | | | Fuzzy | 10017565 |
| | | | | Fuzzy head | 10017566 |
| | | | | Muzzy head | 10028405 |
| | | | | Neck strange feeling | 10028844 |
| | | | | of | |
| | | | | Soft feeling | 10041286 |
| | | | | Spaced out | 10041374 |
| | | | | Thick head | 10043428 |
| | | | | Unstable feeling | 10046253 |
| | | | | Weird feeling | 10047904 |

The AE term of sedation is mentioned in the 2010 Draft Guidance but is not included in this table.

## 10.2 Appendix 2: Drug Withdrawal Related Adverse Events

Drug Withdrawal – Related Adverse Events Occurring Following Drug Discontinuation (Preferred Terms; MedDRA 20.0)

| System Organ<br>Class | Higher Level GT | Higher Level<br>Term | Preferred Term | Preferred Term<br>Code |
|---|---|---|---|---|
| Psychiatric disorders | Anxiety disorders and symptoms | Anxiety symptoms | Agitation | 10001497 |
| Nervous system disorders | Neurological<br>disorders NEC | Neurological signs and symptoms NEC | | 10001497 |
| Psychiatric disorders | Depressed mood disorders and disturbances | Mood alterations with depressive symptoms | Anhedonia | 10002511 |
| Psychiatric disorders | Anxiety disorders and symptoms | Anxiety symptoms | Anxiety | 10002855 |
| Musculoskeletal<br>and connective<br>tissue disorders | Muscle disorders | Muscle related<br>signs and symptoms<br>NEC | Chills | 10008531 |
| Musculoskeletal and connective tissue disorders | Muscle disorders | Feelings and sensations NEC | | 10008531 |
| Psychiatric disorders | Depressed mood disorders and disturbances | Mood alterations with depressive symptoms | Depressed mood | 10012374 |
| Psychiatric disorders | Depressed mood disorders and disturbances | Depressive disorders | Depression | 10012378 |
| Gastrointestinal disorders | Gastrointestinal motility and defaecation conditions | Diarrhoea (excl infective) | Diarrhoea | 10012735 |
| Psychiatric disorders | Mood disorders and disturbances | Emotional and mood disturbances NEC | Dysphoria | 10013954 |
| Nervous system disorders | Sleep disturbances (incl subtypes) | Sleep disturbances<br>NEC | Dyssomnia | 10061827 |
| Psychiatric disorders | Sleep disorders and disturbances | Dyssomnias | | 10061827 |
| Psychiatric disorders | Depressed mood disorders and disturbances | Depressive disorders | Persistent depressive disorder | 10077804 |
| Psychiatric disorders | Depressed mood disorders and disturbances | Mood alterations with depressive symptoms | Feeling of despair | 10016344 |
| Nervous system disorders | Headaches | Headaches NEC | Headache | 10019211 |
| Skin and subcutaneous tissue disorders | Skin appendage conditions | Apocrine and eccrine gland disorders | Hyperhidrosis | 10020642 |
| General disorders<br>and administration<br>site conditions | General system disorders NEC | General signs and symptoms NEC | | 10020642 |
| Psychiatric | Sleep disorders and | Disturbances in | Insomnia | 10022437 |

Gastrointestinal

disorders

| System Organ<br>Class | Higher Level GT | Higher Level<br>Term | Preferred Term | Preferred Term<br>Code |
|---|---|---|---|---|
| disorders | disturbances | initiating and | | Couc |
| uisorucis | disturbances | maintaining sleep | | |
| Nervous system | Sleep disturbances | Disturbances in | - | 10022437 |
| disorders | Sieep disturbances | initiating and | | 10022437 |
| uisolucis | | maintaining sleep | | |
| Psychiatric | Depressed mood | Mood alterations | Morose | 10027977 |
| disorders | disorders and | with depressive | Wiolose | 1002/9// |
| uisoiueis | disturbances | - | | |
| Gastrointestinal | Gastrointestinal | symptoms Nausea and | Nausea | 10020012 |
| | | | Nausea | 10028813 |
| disorders | signs and symptoms | vomiting symptoms | NT (1 1 1) | 10050650 |
| Psychiatric | Depressed mood | Mood alterations | Negative thoughts | 10058672 |
| disorders | disorders and | with depressive | | |
| | disturbances | symptoms | 27 | 100000 |
| Psychiatric | Anxiety disorders | Anxiety symptoms | Nervousness | 10029216 |
| disorders | and symptoms | | | |
| Psychiatric | Anxiety disorders | Obsessive- | Obsessive thoughts | 10029897 |
| disorders | and symptoms | compulsive | | |
| | | disorders and | | |
| | | symptoms | | |
| General disorders | General system | Pain and discomfort | Pain | 10033371 |
| and administration | disorders NEC | NEC | | |
| site conditions | | | | |
| Nervous system | Sleep disturbances | Sleep disturbances | Poor quality sleep | 10062519 |
| disorders | (incl subtypes) | NEC | | |
| Psychiatric | Sleep disorders and | Dyssomnias | | 10062519 |
| disorders | disturbances | | | |
| Cardiac disorders | Cardiac disorder | Cardiac signs and | Syncope | 10042772 |
| | signs and symptoms | symptoms NEC | | |
| Vascular disorders | Decreased and | Circulatory collapse | 1 | 10042772 |
| | nonspecific blood | and shock | | |
| | pressure disorders | | | |
| | and shock | | | |
| Nervous system | Neurological | Disturbances in | - | 10042772 |
| disorders | disorders NEC | consciousness NEC | | -00.2772 |
| Psychiatric | Sleep disorders and | Disturbances in | Terminal insomnia | 10068932 |
| disorders | disturbances | initiating and | (lower level term of | 10000,32 |
| distincts | distait dances | maintaining sleep | interest: early | |
| Nervous system | Sleep disturbances | Disturbances in | morning | 10068932 |
| disorders | Sicep disturbances | initiating and | awakening) | 10000732 |
| uisolucis | | maintaining sleep | awakeming) | |
| Namiona arestone | Mariamant | | Tromor | 10044565 |
| Nervous system | Movement | Tremor (excl | Tremor | 10044565 |
| disorders | disorders (incl | congenital) | | |
| | parkinsonism) | ) · | | 10047700 |

Nausea and

vomiting symptoms

Gastrointestinal

signs and symptoms

Vomiting

10047700

## 10.3 Appendix 3: Potentially Clinically Significant Laboratory Criteria

| Laboratory Parameter | Potentially Clinically Significant Laboratory Criteria | | | | | |
|---|---|---|---|---|---|---|
| Hematology and Coagulation | | Low PCS criteria | High PCS criteria | Conv. | Low PCS criteria | criteria |
| Hemoglobin $< 7.0 \text{ g/L}$ $> 20.0 \text{ g/L}$ $> 200 \text{ g/L}$ $> 200 \text{ g/L}$ Hematocrit $< 20.0 \%$ $> 60.0 \%$ $0.01$ $< 0.200 \text{ v/v}$ (Fraction) $< 0.600 \text{ v/v}$ (Fraction) Leukocytes (White Blood Cell Count) $< 2.00 \times 10^3 / \mu L$ $> 30.00 \times 10^3 / \mu L$ $1$ $< 2.00 \times 10^9 / L$ $> 30.00 \times 10^9 / L$ Platelets $< 40 \times 10^3 / \mu L$ $> 1000 \times 10^3 / \mu L$ $1$ $< 40 \times 10^9 / L$ $> 1000 \times 10^9 / L$ International Normalized Ratio (INR) No lower limit $> 2 \text{ (Ratio)}$ $1$ No lower limit $> 2.00 \text{ (Ratio)}$ Sodium $< 120 \text{ mEq/L}$ $> 160 \text{ mEq/L}$ $1$ $< 120 \text{ mmol/L}$ $> 160 \text{ mmol/L}$ Potassium $< 120 \text{ mEq/L}$ $> 160 \text{ mEq/L}$ $1$ $< 2.8 \text{ mmol/L}$ $> 6.2 \text{ mmol/L}$ Calcium $< 6.0 \text{ mg/dL}$ $> 13.0 \text{ mg/dL}$ $0.25$ $< 1.50 \text{ mmol/L}$ $> 3.25 \text{ mmol/L}$ Magnesium $< 0.98 \text{ mg/dL}$ $> 4.74 \text{ mg/dL}$ $0.4114$ $< 0.400 \text{ mmol/L}$ $> 24.98 \text{ mmol/L}$ Glucose $< 40 \text{ mg/dL}$ $> 450 \text{ mg/dL}$ | | <u> </u> | [amatalogy and Ca | agulation | (Si unit) | (Si unit) |
| Hematocrit | Hamaglahin | | | | < 70 α/I | > 200 a/I |
| $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | Tiemogloom | < 7.0 g/uL | > 20.0 g/uL | 10 | \ 70 g/L | > 200 g/L |
| $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | Hematocrit | < 20 0 % | > 60 0 % | 0.01 | < 0.200 v/v | > 0 600 v/v |
| | 1101114100111 | 20.0 70 | 00.0 70 | 0.01 | | |
| White Blood Cell Count Count Platelets < 40 x10 <sup>3</sup> /μL > 1000 x10 <sup>3</sup> /μL 1 < 40 x10 <sup>9</sup> /L > 1000 x10 <sup>9</sup> /L | Leukocytes | $< 2.00 \text{ x} 10^3 / \mu \text{L}$ | $> 30.00 \text{ x} 10^3/\mu\text{L}$ | 1 | $< 2.00 \text{ x} 10^9 / \text{L}$ | |
| Platelets $< 40 \times 10^3 / \mu L$ $> 1000 \times 10^3 / \mu L$ 1 $< 40 \times 10^9 / L$ $> 1000 \times 10^9 / L$ International Normalized Ratio (INR) No lower limit $> 2$ (Ratio) 1 No lower limit $> 2.00$ (Ratio) Other Biochemistry* Sodium $< 120 \text{ mEq/L}$ $> 160 \text{ mEq/L}$ 1 $< 120 \text{ mmol/L}$ $> 160 \text{ mmol/L}$ Potassium $< 2.8 \text{ mEq/L}$ $> 6.2 \text{ mEq/L}$ 1 $< 2.8 \text{ mmol/L}$ $> 6.2 \text{ mmol/L}$ Calcium $< 6.0 \text{ mg/dL}$ $> 13.0 \text{ mg/dL}$ $0.25$ $< 1.50 \text{ mmol/L}$ $> 3.25 \text{ mmol/L}$ Chloride $< 80 \text{ mEq/L}$ $> 120 \text{ mEq/L}$ 1 $< 80 \text{ mmol/L}$ $> 1.20 \text{ mmol/L}$ Magnesium $< 0.98 \text{ mg/dL}$ $> 4.74 \text{ mg/dL}$ $0.4114$ $< 0.400 \text{ mmol/L}$ $> 1.950 \text{ mmol/L}$ Glucose $< 40 \text{ mg/dL}$ $> 450 \text{ mg/dL}$ $< 0.0555$ $< 2.22 \text{ mmol/L}$ $> 24.98 \text{ mmol/L}$ Creatinine No lower limit $> 5.00 \text{ mg/dL}$ $> 3.48 \text{ No lower limit}$ $> 442.0 \text{ µmol/L}$ Uric Acid No lower limit < | | | · | | | |
| International Normalized Ratio (INR) | Count) | | | | | |
| Normalized Ratio (INR) Other Biochemistry* Sodium < 120 mEq/L | Platelets | $< 40 \text{ x} 10^3 / \mu \text{L}$ | $> 1000 \text{ x} 10^3 / \mu \text{L}$ | 1 | $< 40 \text{ x} 10^9 / \text{L}$ | $> 1000 \text{ x} 10^9 / \text{L}$ |
| Normalized Ratio (INR) Other Biochemistry* Sodium < 120 mEq/L | | | | | | |
| Other Biochemistry* | | No lower limit | > 2 (Ratio) | 1 | No lower limit | > 2.00 (Ratio) |
| Other Biochemistry* Sodium < 120 mEq/L | | | | | | |
| Sodium < 120 mEq/L > 160 mEq/L 1 < 120 mmol/L > 160 mmol/L Potassium < 2.8 mEq/L | (INR) | | O(1 B) 1 : | 4 4 | | |
| Potassium < 2.8 mEq/L > 6.2 mEq/L 1 < 2.8 mmol/L > 6.2 mmol/L Calcium < 6.0 mg/dL | G 1: | 120 E /I | | | . 120 1/I | > 1.60 1/I |
| Calcium < 6.0 mg/dL | Sodium | < 120 mEq/L | > 160 mEq/L | 1 | < 120 mmol/L | > 160 mmol/L |
| Calcium < 6.0 mg/dL | Potaccium | < 2.8 mFa/I | > 6.2 mFa/I | 1 | < 2.8 mmol/I | > 6.2 mmol/I |
| Chloride < 80 mEq/L > 120 mEq/L 1 < 80 mmol/L > 120 mmol/L Magnesium < 0.98 mg/dL | 1 ottassium | 2.0 IIIEq/E | > 0.2 IIIEq/E | 1 | 2.0 mmo/L | > 0.2 mmoi/L |
| Chloride < 80 mEq/L > 120 mEq/L 1 < 80 mmol/L > 120 mmol/L Magnesium < 0.98 mg/dL | Calcium | < 6.0 mg/dL | > 13.0 mg/dL | 0.25 | < 1.50 mmol/L | > 3.25 mmol/L |
| Magnesium < 0.98 mg/dL | | | | | | |
| Glucose $<40 \text{ mg/dL}$ $>450 \text{ mg/dL}$ $0.0555$ $<2.22 \text{ mmol/L}$ $>24.98 \text{ mmol/L}$ Creatinine No lower limit $>5.00 \text{ mg/dL}$ $88.4$ No lower limit $>442.0 \text{ µmol/L}$ Uric Acid No lower limit $>13.0 \text{ mg/dL}$ $59.48$ No lower limit $>773 \text{ µmol/L}$ Blood Urea No lower limit $>80 \text{ mg/dL}$ $0.357$ No lower limit $>28.6 \text{ mmol/L}$ | Chloride | < 80 mEq/L | > 120 mEq/L | 1 | < 80 mmol/L | > 120 mmol/L |
| Glucose $<40 \text{ mg/dL}$ $>450 \text{ mg/dL}$ $0.0555$ $<2.22 \text{ mmol/L}$ $>24.98 \text{ mmol/L}$ Creatinine No lower limit $>5.00 \text{ mg/dL}$ $88.4$ No lower limit $>442.0 \text{ µmol/L}$ Uric Acid No lower limit $>13.0 \text{ mg/dL}$ $59.48$ No lower limit $>773 \text{ µmol/L}$ Blood Urea No lower limit $>80 \text{ mg/dL}$ $0.357$ No lower limit $>28.6 \text{ mmol/L}$ | | | _ | | | |
| Creatinine No lower limit > 5.00 mg/dL 88.4 No lower limit > 442.0 μmol/L Uric Acid No lower limit > 13.0 mg/dL 59.48 No lower limit > 773 μmol/L Blood Urea No lower limit > 80 mg/dL 0.357 No lower limit > 28.6 mmol/L | Magnesium | < 0.98 mg/dL | > 4.74 mg/dL | 0.4114 | < 0.400 mmol/L | > 1.950 mmol/L |
| Creatinine No lower limit > 5.00 mg/dL 88.4 No lower limit > 442.0 μmol/L Uric Acid No lower limit > 13.0 mg/dL 59.48 No lower limit > 773 μmol/L Blood Urea No lower limit > 80 mg/dL 0.357 No lower limit > 28.6 mmol/L | | | | | | |
| Uric Acid No lower limit > 13.0 mg/dL 59.48 No lower limit > 773 μmol/L Blood Urea No lower limit > 80 mg/dL 0.357 No lower limit > 28.6 mmol/L | Glucose | < 40 mg/dL | > 450 mg/dL | 0.0555 | < 2.22 mmol/L | > 24.98 mmol/L |
| Uric Acid No lower limit > 13.0 mg/dL 59.48 No lower limit > 773 μmol/L Blood Urea No lower limit > 80 mg/dL 0.357 No lower limit > 28.6 mmol/L | Q .: : | NT 1 11 11 | . 5.00 /15 | 00.4 | 37 1 11 11 | . 440 O 1/I |
| Blood Urea No lower limit > 80 mg/dL 0.357 No lower limit > 28.6 mmol/L | Creatinine | No lower limit | > 5.00 mg/dL | 88.4 | No lower limit | > 442.0 μmol/L |
| Blood Urea No lower limit > 80 mg/dL 0.357 No lower limit > 28.6 mmol/L | Uric Acid | No lower limit | > 13.0 mg/dI | 50.48 | No lower limit | > 773 umol/I |
| | One Acid | 140 lower millt | - 15.0 mg/uL | 39.40 | 140 lower millit | - //3 μποι/L |
| | Blood Urea | No lower limit | > 80 mg/dL | 0.357 | No lower limit | > 28 6 mmol/L |
| | | 1.0 10 110 1111111 | 00 1119, 412 | 0.557 | 1.0 10 Wel milit | 20.0 1111101112 |
| | (= 0-1) | | | | | |

Source: Tietz. Textbook of Clinical Chemistry and Molecular Diagnostics, 4<sup>th</sup> Edition. Elsevier Saunders, 2006, section VII, chapter 56, pages 2317-2318.

Conv.: Conversion; PCS: Potentially Clinically Significant; SI: International System of Units.

<sup>\*</sup> PCS criteria for Liver Enzymes and Total Bilirubin are provided in Table 22. Section 7.5.3.1

## 10.4 Appendix 4: Key Contributors and Approvers

## **List of Key Contributors and Approvers**

#### **Key Contributors**

The following contributed to or reviewed this Statistical Analysis Plan as relevant to their indicated discipline or role.

| Primary author (s) |
|-----------------------------------|
| M.S., |
| <b>Contributors and Reviewers</b> |
| PhD, Director, |
| MD PhD, |
| PhD, |

## **Author and Approver Signatories**

| Authored by: | | |
|--------------|--------|--------------------|
| | , M.S. | Date (DD Mmm YYYY) |

(E-signatures are attached at end of document)

| Astellas Pharma Global |
|---------------------------------------|
| wer of this Statistical Analysis Plan |

This Statistical Analysis Plan was approved by:

PhD

Astellas Pharma Global Development, Inc.

This Statistical Analysis Plan was approved by:

MD, PhD,

Astellas Pharma Global Development, Inc.